CLINICAL TRIAL: NCT04563845
Title: A Study to Evaluate the Effect of Therapeutic and Supratherapeutic Oral Doses of GSK3640254 on Cardiac Conduction as Assessed by 12-Lead Electrocardiogram Compared to Placebo and a Single Oral Dose of Moxifloxacin in Healthy Adult Participants
Brief Title: Effect of Therapeutic and Supratherapeutic Oral Doses of GSK3640254 on Cardiac Conduction Compared to Placebo and a Single Oral Dose of Moxifloxacin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 213053
Record Dates: First submitted 2020-09-18; First posted 2020-09-25 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: HIV Infections
Keywords: GSK3640254; Moxifloxacin; Electrocardiogram; Cardiac Conduction; Supratherapeutic dose
MeSH Terms: conditions — HIV Infections | interventions — GSK3640254; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Participants receiving placebo (Placebo Comparator): Participants will receive a single dose of placebo once daily for 7 days following ingestion of a moderate fat meal.
  Interventions: Drug: GSK3640254; Drug: Placebo
- Part 1: Participants receiving GSK3640254 500 milligrams (mg) (Experimental): Participants will receive a single dose of GSK3640254 500 mg once daily for 7 days following ingestion of a moderate fat meal.
  Interventions: Drug: GSK3640254
- Part 2: Main QTc Study (Experimental): Participants will be randomized to 1:1:1:1 ratio to receive Treatment T- Therapeutic dose of GSK3640254 (100 mg QD) on Days 1 through 7 or Treatment ST- Supratherapeutic dose of GSK3640254 (to be determined from Part 1) on Days 1 through 7 or Treatment P- Placebo for GSK3640254 on Days 1 through 7 or Treatment M- Moxifloxacin (GSK3640254 placebo Days 1 through 6 and a single dose of Moxifloxacin [400 mg] on Day 7 in 4 treatment periods. There will be at least 7 days wash out period between each period.
  Interventions: Drug: GSK3640254; Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: GSK3640254 — GSK3640254 will be administered.
Drug: Placebo — Placebo will be administered.
  Arms: Part 1: Participants receiving placebo; Part 2: Main QTc Study
Drug: Moxifloxacin — Moxifloxacin will be administered.
  Arms: Part 2: Main QTc Study

SUMMARY:
This study will aim to evaluate the effect of therapeutic and supratherapeutic oral doses of GSK3640254 on cardiac conduction compared to placebo and a single oral dose of Moxifloxacin in healthy adult participants. The study has 2 parts: Part 1 will determine the supratherapeutic dose for Part 2, which will be the main corrected QT interval (QTc) study. Part 1 will evaluate once daily (QD) dosing of GSK3640254 or placebo and Part 2 will investigate the safety, tolerability and Pharmacokinetics (PK) of GSK3640254 doses on cardiac conduction as compared to placebo and a single oral dose of Moxifloxacin in healthy adult participants. Moxifloxacin will be included as a positive control.

ELIGIBILITY:
Inclusion criteria:

* Participant must be 18 to 50 years of age inclusive, at the time of signing the informed consent.
* Participants who are healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination (including cardiopulmonary examination), laboratory tests, and cardiac monitoring (history and ECG).
* Body weight more than or equal to (>=)50.0 kilograms (kg) (110 pounds [lbs]) for men and >=45.0 kg (99 lbs) for women and body mass index within the range 18.5 to 31.0 kilograms per square meter (kg/m^2) (inclusive).
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Male or female participants:

  1. Male participants should not engage in intercourse while confined in the clinic. There is no need for an extended period of double barrier use or prolonged abstinence after study discharge.
  2. Female participants:

  (i) A female participant is eligible to participate if she is not pregnant, planning to become pregnant within the next 6 months, or breastfeeding, and at least 1 of the following conditions applies: Is not a woman of childbearing potential (WOCBP) OR Is a WOCBP and using a non-hormonal contraceptive method that is highly effective, with a failure rate of less than (<)1 percent (%) for 28 days before intervention, during the intervention period, and for at least 28 days after the last dose of study intervention. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

(ii) A WOCBP must have a negative highly sensitive serum pregnancy test at Screening and Check-in.

* Capable of giving signed informed, which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and in this protocol.

Exclusion criteria:

* Participants with current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A pre-existing condition interfering with normal Gastrointestinal (GI) anatomy or motility (for example [e.g.], gastro-esophageal reflux disease, gastric ulcers, gastritis), hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study intervention or render the participant unable to take oral study intervention.
* Prior cholecystectomy (prior appendectomy is acceptable).
* Clinically significant illness, including viral syndromes, within 3 weeks of dosing.
* A participant with known or suspected active Coronavirus Disease-2019 (COVID-19) infection OR contact with an individual with known COVID-19, within 14 days of study enrollment (World Health Organization [WHO] definitions).
* Any history of significant underlying psychiatric disorder, including, but not limited to, schizophrenia, bipolar disorder with or without psychotic symptoms, other psychotic disorders, or schizotypal (personality) disorder.
* Any history of major depressive disorder with or without suicidal features, or anxiety disorders that required medical intervention (pharmacologic or not) such as hospitalization or other inpatient treatment and/or chronic (more than [>]6 months) outpatient treatment. Participants with other conditions such as adjustment disorder or dysthymia that have required shorter term medical therapy (<6 months) without inpatient treatment and are currently well-controlled clinically or resolved may be considered for entry after discussion and agreement with the ViiV Healthcare/GlaxoSmithKline (VH/GSK) Medical Monitor.
* Any pre-existing physical or other psychiatric condition (including alcohol or drug abuse), which, in the opinion of the investigator (with or without psychiatric evaluation), could interfere with the participant's ability to comply with the dosing schedule and protocol evaluations or which might compromise the safety of the participant.
* Medical history of cardiac arrhythmias, prior myocardial infarction in the past 3 months, or cardiac disease or a family or personal history of long QT syndrome.
* History indicative of an increased risk of a cardiac arrhythmia or cardiac disease, including the following:

  1. History of symptomatic cardiac arrhythmias or palpitations associated with pre-syncope or syncope, or history of unexplained syncope.
  2. History of cardiac arrest.
  3. History of clinically relevant cardiac disease including symptomatic or asymptomatic arrhythmias (including but not limited to ventricular fibrillation, ventricular tachycardia, any degree of atrioventricular block, Brugada syndrome, Wolff-Parkinson-White Syndrome, and sinus bradycardia, defined as HR less than 50 bpm based on vital signs or ECG), presyncope or syncopal episodes, or additional risk factors for torsades de pointes (e.g., heart failure).
  4. History of clinically relevant structural cardiac disease including hypertrophic obstructive cardiomyopathy.
  5. History of hypokalemia.
* History of heart disease (e.g., coronary heart disease, angina).
* Presence of hepatitis B surface antigen at Screening or within 3 months prior to starting study intervention.
* Positive hepatitis C antibody test result at Screening or within 3 months prior to starting study intervention.
* Positive Human Immunodeficiency virus (HIV)-1 and -2 antigen/antibody immunoassay at Screening.
* Alanine aminotransferase (ALT) >=1.5 times upper limit of normal (ULN). A single repeat of ALT is allowed within a single Screening period to determine eligibility.
* Bilirubin >=1.5 times ULN (isolated bilirubin >=1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat of any laboratory abnormality is allowed within a single Screening period to determine eligibility.
* Any acute laboratory abnormality (including hypokalemia, hypercalcemia, or hypomagnesemia) at Screening which, in the opinion of the investigator, should preclude participation in the study of an investigational compound.
* Any Grade 2 to 4 laboratory abnormality at Screening, with the exception of lipid abnormalities (e.g., total cholesterol, triglycerides), and ALT (previously described), will exclude a participant from the study unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the sponsor. A single repeat of any laboratory abnormality is allowed within a single Screening period to determine eligibility.
* Urine drug screen positive (showing presence of): amphetamines, barbiturates, cocaine, Methylenedioxymethamphetamine (MDMA), cannabinoids, methamphetamines, phencyclidine, or non-prescribed opiates, oxycodone, benzodiazepines, methadone, or tricyclic antidepressants at screening or before dosing of study intervention.
* Unable to refrain from the use of prescription or nonprescription drugs including vitamins, herbal and dietary supplements (including Saint [St] John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study intervention and for the duration of the study.
* Treatment with any vaccine within 30 days prior to receiving study intervention.
* Unwillingness to abstain from consumption of any food or drink containing grapefruit and grapefruit juice, Seville oranges, blood oranges, or pomelos or their fruit juices within 7 days prior to the first dose of study intervention(s) until the end of the study.
* Participation in another concurrent clinical study or prior clinical study (with the exception of imaging trials) prior to the first dosing day in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the study intervention (whichever is longer).
* Prior exposure to GSK3640254 in this or another clinical study.
* Prior intolerance to Moxifloxacin.
* Prior participation in this clinical study (participants may not participate in both Part 1 and Part 2 of the study).
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* Any positive (abnormal) response confirmed by the investigator on a screening clinician- or qualified designee-administered Columbia-Suicide Severity Rating Scale (C-SSRS).
* A sustained supine systolic blood pressure >150 millimeters of mercury (mm Hg) or <90 mm Hg or a supine diastolic blood pressure >95 mm Hg or <50 mm Hg at Screening or Check-in (Day -2). Blood pressure may be retested once in the supine position. The blood pressure abnormality is considered sustained if either the systolic or the diastolic pressure values are outside the stated limits after 2 assessments, in which case the participant may not be randomized.
* A resting HR of <50 bpm or >100 bpm when vital signs are measured at Screening or Check-in (Day -2). A HR from 100 to 110 bpm can be rechecked by ECG or vital signs within up to 2 hours to verify eligibility.
* An uninterpretable ECG or any significant arrhythmia or ECG finding (e.g., prior myocardial infarction in the past 3 months, significant pathological Q-waves (defined as Q-wave >40 ms or depth greater than 0.4-0.5 millivolts [mV], symptomatic bradycardia, non-sustained or sustained atrial arrhythmias, ventricular pre-excitation, non-sustained or sustained ventricular tachycardia, any degree of atrioventricular block, complete left bundle branch block, or conduction abnormality) which, in the opinion of the investigator or VH/GSK Medical Monitor, will interfere with the safety of the individual participant.
* Exclusion criteria for Screening ECG (a single repeat is allowed for eligibility determination):

  (i) HR: <50 or >100 bpm (ii) QTcF interval1: >450 ms (iii) QRS interval: >110 ms (iv) PR interval: >200 ms
* Screening Holter (24 hours) with any of the following:

  (i) Sinus bradycardia less than or equal to (<=)35 bpm or junctional arrhythmia >60 bpm for 10 seconds or longer.

(ii) Non-sustained ventricular tachycardia or more than 30 ventricular premature depolarizations during an hour.

(iii) Atrial arrhythmia >100 bpm for 3 seconds or longer or more than 40 atrial premature depolarizations during an hour.

* History of alcoholism and/or drug/chemical abuse or regular alcohol consumption within 6 months of screening, defined as an average weekly intake of >14 units. One unit is equivalent to 8 grams of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine, or 1 (25 mL) measure of spirits.
* Unable to refrain from tobacco or nicotine-containing products within 3 months prior to Screening and for the duration of the study.
* History of sensitivity to any of the study medications or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Zhang Y, Bush M, Yazdani P, Zhan J, Wen B, Bainbridge V, Wynne BR, Joshi S, Lataillade M. Effects of the HIV-1 maturation inhibitor GSK3640254 on QT interval in healthy participants. Pharmacol Res Perspect. 2023 Dec;11(6):e01151. doi: 10.1002/prp2.1151. PMID 37961928

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States.
Pre-assignment Details: A total of 50 participants (8 in Part 1 and 42 in Part 2) were enrolled in the study (Safety Population: It comprised of all participants who received at least 1 dose of study intervention).
Groups:
- Part 1: Placebo: Participants received a single dose of placebo once daily for 7 days following ingestion of a moderate fat meal.
- Part 1: GSK3640254 500 mg: Participants received single dose of GSK3640254 500 mg once daily for 7 days following ingestion of a moderate fat meal.
- Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg: Participants received a single therapeutic dose of GSK3640254 100 mg once daily on Days 1 through 7 (Treatment T) in treatment period 1. In treatment period 2, participants received single supratherapeutic dose of GSK3640254 500 mg once daily on Days 1 through 7 (Treatment ST). In treatment period 3, participants received placebo for GSK3640254 on Days 1 through 7 (Treatment P). In treatment period 4, participants received placebo for GSK3640254 on Days 1 through 6 and a single dose of moxifloxacin 400 mg on Day 7 (Treatment M). There was a washout period of at least 7 days between each treatment periods.
- Part 2: GSK3640254 500 mg/Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo: Participants received single supratherapeutic dose of GSK3640254 500 mg on Days 1 through 7 (Treatment ST) in treatment period 1. In treatment period 2, participants received placebo for GSK3640254 on Days 1 through 6 and a single dose of moxifloxacin 400 mg on Day 7 (Treatment M). In treatment period 3, participants received a single therapeutic dose of GSK3640254 100 mg on Days 1 through 7 (Treatment T). In treatment period 4, participants received placebo for GSK3640254 on Days 1 through 7 (Treatment P). There was a washout period of at least 7 days between each treatment periods.
- Part 2: Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg/GSK3640254 500 mg: Participants received placebo for GSK3640254 on Days 1 through 7 (Treatment P) in treatment period 1. In treatment period 2, participants received a single therapeutic dose of GSK3640254 100 mg on Days 1 through 7 (Treatment T). In treatment period 3, participants received placebo for GSK3640254 on Days 1 through 6 and a single dose of moxifloxacin 400 mg on Day 7 (Treatment M). In treatment period 4, participants received single supratherapeutic dose of GSK3640254 500 mg on Days 1 through 7 (Treatment ST). There was a washout period of at least 7 days between each treatment periods.
- Part 2: Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg/GSK3640254 100 mg: Participants received placebo for GSK3640254 on Days 1 through 6 and a single dose of moxifloxacin 400 mg on Day 7 (Treatment M) in treatment period 1. In treatment period 2, participants received placebo for GSK3640254 on Days 1 through 7 (Treatment P). In treatment period 3, participants received single supratherapeutic dose of GSK3640254 500 mg on Days 1 through 7 (Treatment ST). In treatment period 4, participants received a single therapeutic dose of GSK3640254 100 mg on Days 1 through 7 (Treatment T). There was a washout period of at least 7 days between each treatment periods.
- Part 2: GSK3640254 500 mg/Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg: Participants received single supratherapeutic dose of GSK3640254 500 mg on Days 1 through 7 (Treatment ST) in treatment period 1. In treatment period 2, participants received placebo for GSK3640254 on Days 1 through 7 (Treatment P). In treatment period 3, participants received a single therapeutic dose of GSK3640254 100 mg on Days 1 through 7 (Treatment T). In treatment period 4, participants received placebo for GSK3640254 on Days 1 through 6 and a single dose of moxifloxacin 400 mg on Day 7(Treatment M). There was a washout period of at least 7 days between each treatment periods.
- Part 2: Placebo/Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg: Participants received placebo for GSK3640254 on Days 1 through 7 (Treatment P) in treatment period 1. In treatment period 2, participants received placebo for GSK3640254 on Days 1 through 6 and a single dose of moxifloxacin 400 mg on Day 7 (Treatment M). In treatment period 3, participants received single supratherapeutic dose of GSK3640254 500 mg on Days 1 through 7 (Treatment ST). In treatment period 4, participants received a single therapeutic dose of GSK3640254 100 mg on Days 1 through 7 (Treatment T). There was a washout period of at least 7 days between each treatment periods.
- Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg/ Placebo: Participants received a single therapeutic dose of GSK3640254 100 mg Days 1 through 7 (Treatment T) in treatment period 1. In treatment period 2, participants received single supratherapeutic dose of GSK3640254 500 mg Days 1 through 7 (Treatment ST). In treatment period 3, participants received placebo for GSK3640254 on Days 1 through 6 and a single dose of moxifloxacin 400 mg on Day 7 (Treatment M). In treatment period 4, participants received placebo for GSK3640254 on Days 1 through 7 (Treatment P). There was a washout period of at least 7 days between each treatment periods.
- Part 2: Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo/GSK3640254 500 mg: Participants received placebo for GSK3640254 on Days 1 through 6 and a single dose of moxifloxacin 400 mg on Day 7 (Treatment M) in treatment period 1. In treatment period 2, participants received a single therapeutic dose of GSK3640254 100 mg on Days 1 through 7 (Treatment T). In treatment period 3, participants received placebo for GSK3640254 on Days 1 through 7 (Treatment P). In treatment period 4, participants received single supratherapeutic dose of GSK3640254 500 mg on Days 1 through 7 (Treatment ST). There was a washout period of at least 7 days between each treatment periods.
- Part 2: Placebo/GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg: Participants received placebo for GSK3640254 on Days 1 through 7 (Treatment P) in treatment period 1. In treatment period 2, participants received a single therapeutic dose of GSK3640254 100 mg on Days 1 through 7 (Treatment T). In treatment period 3, participants received single supratherapeutic dose of GSK3640254 500 mg on Days 1 through 7 (Treatment ST). In treatment period 4, participants received placebo for GSK3640254 on Days 1 through 6 and a single dose of moxifloxacin 400 mg on Day 7 (Treatment M). There was a washout period of at least 7 days between each treatment periods.
- Part 2: GSK3640254 100 mg/Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg: Participants received a single therapeutic dose of GSK3640254 100 mg on Days 1 through 7 (Treatment T) in treatment period 1. In treatment period 2, participants received placebo for GSK3640254 on Days 1 through 6 and a single dose of moxifloxacin 400 mg on Day 7 (Treatment M). In treatment period 3, participants received placebo for GSK3640254 on Days 1 through 7 (Treatment P). In treatment period 4, participants received single supratherapeutic dose of GSK3640254 500 mg Days 1 through 7 (Treatment ST). There was a washout period of at least 7 days between each treatment periods.
- Part 2: GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg/GSK3640254 100 mg: Participants received single supratherapeutic dose of GSK3640254 500 mg Days 1 through 7 (Treatment ST) in treatment period 1. In treatment period 2, participants received placebo for GSK3640254 on Days 1 through 7 (Treatment P). In treatment period 3, participants received placebo for GSK3640254 on Days 1 through 6 and a single dose of moxifloxacin 400 mg on Day 7 (Treatment M). In treatment period 4, participants received a single therapeutic dose of GSK3640254 100 mg on Days 1 through 7 (Treatment T). There was a washout period of at least 7 days between each treatment periods.
- Part 2: Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg/Placebo: Participants received placebo for GSK3640254 on Days 1 through 6 and a single dose of moxifloxacin 400 mg on Day 7 (Treatment M) in treatment period 1. In treatment period 2, participants received single supratherapeutic dose of GSK3640254 500 mg on Days 1 through 7 (Treatment ST). In treatment period 3, participants received a single therapeutic dose of GSK3640254 100 mg on Days 1 through 7 (Treatment T). In treatment period 4, participants received placebo for GSK3640254 on Days 1 through 7 (Treatment P). There was a washout period of at least 7 days between each treatment periods.
Period: Part 1: (Up to Day 9)
Arm/Group | Part 1: Placebo | Part 1: GSK3640254 500 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg | Part 2: GSK3640254 500 mg/Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo | Part 2: Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg/GSK3640254 500 mg | Part 2: Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 500 mg/Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg | Part 2: Placebo/Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg/ Placebo | Part 2: Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo/GSK3640254 500 mg | Part 2: Placebo/GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg/Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg | Part 2: GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg/GSK3640254 100 mg | Part 2: Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg/Placebo
Started | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2:Treatment Period 1(Up to 7 Days)
Arm/Group | Part 1: Placebo | Part 1: GSK3640254 500 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg | Part 2: GSK3640254 500 mg/Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo | Part 2: Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg/GSK3640254 500 mg | Part 2: Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 500 mg/Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg | Part 2: Placebo/Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg/ Placebo | Part 2: Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo/GSK3640254 500 mg | Part 2: Placebo/GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg/Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg | Part 2: GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg/GSK3640254 100 mg | Part 2: Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg/Placebo
Started | 0 | 0 | 3 | 4 | 4 | 4 | 4 | 3 | 3 | 3 | 4 | 4 | 3 | 3
Completed | 0 | 0 | 3 | 4 | 4 | 4 | 4 | 2 | 3 | 3 | 4 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2:Washout Period 1(Up to 7 Days)
Arm/Group | Part 1: Placebo | Part 1: GSK3640254 500 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg | Part 2: GSK3640254 500 mg/Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo | Part 2: Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg/GSK3640254 500 mg | Part 2: Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 500 mg/Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg | Part 2: Placebo/Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg/ Placebo | Part 2: Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo/GSK3640254 500 mg | Part 2: Placebo/GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg/Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg | Part 2: GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg/GSK3640254 100 mg | Part 2: Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg/Placebo
Started | 0 | 0 | 3 | 4 | 4 | 4 | 4 | 2 | 3 | 3 | 4 | 4 | 3 | 3
Completed | 0 | 0 | 3 | 4 | 3 | 4 | 4 | 2 | 3 | 3 | 4 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2:Treatment Period 2(Up to 7 Days)
Arm/Group | Part 1: Placebo | Part 1: GSK3640254 500 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg | Part 2: GSK3640254 500 mg/Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo | Part 2: Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg/GSK3640254 500 mg | Part 2: Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 500 mg/Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg | Part 2: Placebo/Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg/ Placebo | Part 2: Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo/GSK3640254 500 mg | Part 2: Placebo/GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg/Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg | Part 2: GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg/GSK3640254 100 mg | Part 2: Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg/Placebo
Started | 0 | 0 | 3 | 4 | 3 | 4 | 4 | 2 | 3 | 3 | 4 | 4 | 3 | 3
Completed | 0 | 0 | 3 | 4 | 3 | 4 | 4 | 2 | 3 | 3 | 4 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2:Washout Period 2(Up to 7 Days)
Arm/Group | Part 1: Placebo | Part 1: GSK3640254 500 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg | Part 2: GSK3640254 500 mg/Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo | Part 2: Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg/GSK3640254 500 mg | Part 2: Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 500 mg/Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg | Part 2: Placebo/Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg/ Placebo | Part 2: Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo/GSK3640254 500 mg | Part 2: Placebo/GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg/Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg | Part 2: GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg/GSK3640254 100 mg | Part 2: Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg/Placebo
Started | 0 | 0 | 3 | 4 | 3 | 4 | 4 | 2 | 3 | 3 | 4 | 4 | 3 | 3
Completed | 0 | 0 | 3 | 4 | 3 | 4 | 4 | 2 | 3 | 3 | 4 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2:Treatment Period 3(Up to 7 Days)
Arm/Group | Part 1: Placebo | Part 1: GSK3640254 500 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg | Part 2: GSK3640254 500 mg/Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo | Part 2: Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg/GSK3640254 500 mg | Part 2: Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 500 mg/Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg | Part 2: Placebo/Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg/ Placebo | Part 2: Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo/GSK3640254 500 mg | Part 2: Placebo/GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg/Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg | Part 2: GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg/GSK3640254 100 mg | Part 2: Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg/Placebo
Started | 0 | 0 | 3 | 4 | 3 | 4 | 4 | 2 | 3 | 3 | 4 | 4 | 3 | 3
Completed | 0 | 0 | 3 | 4 | 3 | 4 | 4 | 2 | 3 | 3 | 4 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2:Washout Period 3(Up to 7 Days)
Arm/Group | Part 1: Placebo | Part 1: GSK3640254 500 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg | Part 2: GSK3640254 500 mg/Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo | Part 2: Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg/GSK3640254 500 mg | Part 2: Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 500 mg/Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg | Part 2: Placebo/Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg/ Placebo | Part 2: Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo/GSK3640254 500 mg | Part 2: Placebo/GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg/Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg | Part 2: GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg/GSK3640254 100 mg | Part 2: Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg/Placebo
Started | 0 | 0 | 3 | 4 | 3 | 4 | 4 | 2 | 3 | 3 | 4 | 4 | 3 | 3
Completed | 0 | 0 | 3 | 4 | 3 | 4 | 4 | 2 | 3 | 3 | 4 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2:Treatment Period 4(Up to 7 Days)
Arm/Group | Part 1: Placebo | Part 1: GSK3640254 500 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg | Part 2: GSK3640254 500 mg/Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo | Part 2: Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg/GSK3640254 500 mg | Part 2: Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 500 mg/Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg | Part 2: Placebo/Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg/ Placebo | Part 2: Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo/GSK3640254 500 mg | Part 2: Placebo/GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg/Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg | Part 2: GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg/GSK3640254 100 mg | Part 2: Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg/Placebo
Started | 0 | 0 | 3 | 4 | 3 | 4 | 4 | 2 | 3 | 3 | 4 | 4 | 3 | 3
Completed | 0 | 0 | 3 | 4 | 3 | 4 | 4 | 2 | 3 | 3 | 4 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: GSK3640254 500 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg | Part 2: GSK3640254 500 mg/Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo | Part 2: Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg/GSK3640254 500 mg | Part 2: Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 500 mg/Placebo/GSK3640254 100 mg/Moxifloxacin 400 mg | Part 2: Placebo/Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg | Part 2: GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg/ Placebo | Part 2: Moxifloxacin 400 mg/GSK3640254 100 mg/Placebo/GSK3640254 500 mg | Part 2: Placebo/GSK3640254 100 mg/GSK3640254 500 mg/Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg/Moxifloxacin 400 mg/Placebo/GSK3640254 500 mg | Part 2: GSK3640254 500 mg/Placebo/Moxifloxacin 400 mg/GSK3640254 100 mg | Part 2: Moxifloxacin 400 mg/GSK3640254 500 mg/GSK3640254 100 mg/Placebo | Total
Number analyzed (Participants) | 2 | 6 | 3 | 4 | 4 | 4 | 4 | 3 | 3 | 3 | 4 | 4 | 3 | 3 | 50
Age, Customized [Count of Participants; unit: Participants]
  18-50 years | 2 | 6 | 3 | 4 | 4 | 4 | 4 | 3 | 3 | 3 | 4 | 4 | 3 | 3 | 50
  >50 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 15
  Male | 2 | 2 | 2 | 4 | 1 | 3 | 4 | 3 | 2 | 2 | 1 | 3 | 3 | 3 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-Central/South Asian Heritage | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 1 | 2 | 0 | 1 | 2 | 2 | 1 | 2 | 3 | 0 | 1 | 1 | 2 | 2 | 20
  Native Hawaiian or other pacific islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 1 | 4 | 3 | 2 | 2 | 2 | 3 | 1 | 0 | 3 | 2 | 3 | 1 | 1 | 28

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Plasma Concentration-time Curve From Time Zero to Time t (AUC[0-t]) of GSK3640254
Description: Blood samples were collected at indicated time points. Pharmacokinetic (PK) analysis was conducted using standard non-compartmental methods.
Time Frame: Pre-dose and 30 minutes, 1 Hour, 2 Hours, 3 Hours, 3 Hours 30 minutes, 4 Hours, 4 Hours 30 minutes, 5 Hours, 6 Hours, 12 Hours, 24 Hours, 48 Hours post-dose on Day 7
Population: Pharmacokinetic Parameter Population comprised of all participants who undergone plasma PK sampling and had evaluable PK parameters estimated. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 1: GSK3640254 500 mg
Number analyzed (Participants) | 6
Hours*nanograms per milliliter | 102400 (25.3)

2. Primary Outcome: Part 1: AUC From Time Zero to the End of the Dosing Interval at Steady State (AUC[0-tau]) of GSK3640254
Description: Blood samples were collected at indicated time points. PK analysis was conducted using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: Pharmacokinetic Parameter Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 1: GSK3640254 500 mg
Number analyzed (Participants) | 6
Hours*nanograms per milliliter | 68790 (25.1)

3. Primary Outcome: Part 1: Maximum Observed Concentration (Cmax) of GSK3640254
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1: GSK3640254 500 mg
Number analyzed (Participants) | 6
Nanograms per milliliter | 4439 (22.7)

4. Primary Outcome: Part 1: Plasma Concentration at the End of the Dosing Interval (Ctau) of GSK3640254
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1: GSK3640254 500 mg
Number analyzed (Participants) | 6
Nanograms per milliliter | 2081 (32.4)

5. Primary Outcome: Part 1: Time of Maximum Observed Concentration (Tmax) of GSK3640254
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK3640254 500 mg
Number analyzed (Participants) | 6
Hours | 4.500 [2.00 to 4.50]

6. Primary Outcome: Part 1: Plasma Concentration of GSK3640254
Description: Blood samples were collected at indicated time points to analyze the plasma concentration of GSK3640254.
Time Frame: Pre-dose and 30 minutes, 1 Hour, 2 Hour, 3 Hours, 3 Hours 30 minutes, 4 Hours, 4 Hours 30 minutes, 5 Hours, 6 Hours, 12 Hours, 24 Hours, 48 Hours post-dose on Day 7
Population: Pharmacokinetic concentration Population comprised of all participants who undergone plasma PK sampling and had evaluable PK assay results. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Part 1: GSK3640254 500 mg
Number analyzed (Participants) | 6
Nanograms per milliliter
  Pre-dose, Day 7 | 2168 (668.17)
  30 minutes, Day 7 | 2000 (638.53)
  1 Hour, Day 7 | 2579 (972.02)
  2 Hour, Day 7 | 3513 (1297.2)
  3 Hour, Day 7 | 4228 (997.39)
  3 Hours 30 minutes, Day 7 | 4155 (1042.5)
  4 Hour, Day 7 | 4213 (921.36)
  4 Hours 30 minutes, Day 7 | 4452 (916.01)
  5 Hour, Day 7 | 3840 (1299.8)
  6 Hour, Day 7 | 4010 (934.73)
  12 Hour, Day 7 | 2773 (535.66)
  24 Hour, Day 7 | 2115 (640.77)
  48 Hour, Day 7 | 1070 (412.36)

7. Primary Outcome: Part 1: Plasma Concentration of Major Metabolites of GSK3640254
Description: Blood samples were to be collected at indicated time points to analyze the plasma concentration of major metabolites of GSK3640254.
Time Frame: as for outcome 6
Population: Pharmacokinetic concentration Population. Data was not collected for metabolites of GSK3640254 as there were not enough residual plasma left to analyze metabolites.
Arm/Group | Part 1: GSK3640254 500 mg
Number analyzed (Participants) | 0

8. Primary Outcome: Part 1: Number of Participants With Serious Adverse Events (SAEs) and Non-SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect as per medical and scientific judgment. Adverse events which were not Serious Adverse Events were considered as Non-Serious adverse events.
Time Frame: Up to Day 9
Population: Safety Population comprised of all randomized participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 : Placebo: Participants received a single dose of placebo once daily for 7 days following ingestion of a moderate fat meal.
- Part 1 : GSK3640254 500 mg: Participants received single dose of GSK3640254 500 mg once daily for 7 days following ingestion of a moderate fat meal.
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Participants
  Non SAE | 2 | 1
  SAE | 0 | 0

9. Primary Outcome: Part 1: Absolute Values for Hematology Parameter: Hemoglobin
Description: Blood samples were collected at indicated time points to analyze hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Grams per liter
  Baseline (Day -2) | 143.5 (9.19) | 131.8 (15.65)
  Day 3 | 149.5 (3.54) | 137.3 (15.81)
  Day 7 | 151.5 (2.12) | 140.5 (18.51)
  Day 9 | 152.0 (7.07) | 137.7 (15.82)

10. Primary Outcome: Part 1: Absolute Values for Hematology Parameter: Hematocrit
Description: Blood samples were collected at indicated time points to analyze hematocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Proportion of red blood cells in blood
  Baseline (Day -2) | 0.4155 (0.03041) | 0.3920 (0.03663)
  Day 3 | 0.4365 (0.00636) | 0.4048 (0.03596)
  Day 7 | 0.4405 (0.00636) | 0.4140 (0.04358)
  Day 9 | 0.4465 (0.01626) | 0.4062 (0.03896)

11. Primary Outcome: Part 1: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected at indicated time points to analyze erythrocytes mean corpuscular volume. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Median (Standard Deviation); unit: Femtoliter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Femtoliter
  Baseline (Day -2) | 87.70 (7.920) | 84.42 (5.398)
  Day 3 | 87.30 (7.071) | 83.95 (5.315)
  Day 7 | 87.30 (7.637) | 84.05 (4.980)
  Day 9 | 88.20 (7.495) | 83.67 (4.815)

12. Primary Outcome: Part 1: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected at indicated time points to analyze erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Picograms
  Baseline (Day-2) | 30.35 (2.475) | 28.35 (2.299)
  Day 3 | 29.85 (2.616) | 28.43 (2.417)
  Day 7 | 30.00 (2.546) | 28.50 (2.269)
  Day 9 | 30.00 (2.828) | 28.33 (2.087)

13. Primary Outcome: Part 1: Absolute Values for Hematology Parameter: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets and Leukocytes
Description: Blood samples were collected at indicated time points to analyze basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelets and leukocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. .
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
10^9 cells per liter
  Basophils, Baseline (Day -2) | 0.070 (0.0424) | 0.057 (0.0163)
  Basophils, Day 3 | 0.065 (0.0212) | 0.053 (0.0186)
  Basophils, Day 7 | 0.065 (0.0212) | 0.048 (0.0160)
  Basophils, Day 9 | 0.060 (0.0000) | 0.065 (0.0176)
  Eosinophils, Baseline (Day -2) | 0.375 (0.0071) | 0.137 (0.1166)
  Eosinophils, Day 3 | 0.350 (0.1838) | 0.115 (0.0794)
  Eosinophils, Day 7 | 0.345 (0.2758) | 0.102 (0.0804)
  Eosinophils, Day 9 | 0.330 (0.2546) | 0.097 (0.0833)
  Lymphocytes, Baseline (Day -2) | 2.520 (0.2828) | 1.822 (0.6201)
  Lymphocytes, Day 3 | 2.715 (0.5020) | 1.657 (0.5352)
  Lymphocytes, Day 7 | 2.515 (0.1202) | 1.668 (0.5780)
  Lymphocytes, Day 9 | 2.100 (0.0990) | 1.935 (0.7973)
  Monocytes, Baseline (Day -2) | 0.550 (0.1414) | 0.537 (0.1878)
  Monocytes, Day 3 | 0.570 (0.1980) | 0.462 (0.1253)
  Monocytes, Day 7 | 0.525 (0.0919) | 0.490 (0.1685)
  Monocytes, Day 9 | 0.490 (0.1980) | 0.508 (0.1411)
  Neutrophils, Baseline (Day -2) | 4.010 (3.3375) | 3.910 (0.4029)
  Neutrophils, Day 3 | 4.300 (3.8608) | 3.015 (1.0263)
  Neutrophils, Day 7 | 4.205 (3.6557) | 3.278 (0.8286)
  Neutrophils, Day 9 | 5.215 (5.1831) | 3.168 (0.8168)
  Platelets, Baseline (Day -2) | 228.0 (50.91) | 266.5 (83.32)
  Platelets, Day 3 | 233.0 (59.40) | 264.2 (75.68)
  Platelets, Day 7 | 243.5 (68.59) | 280.0 (72.09)
  Platelets, Day 9 | 239.0 (82.02) | 269.8 (74.88)
  Leukocytes, Baseline (Day -2) | 7.35 (3.606) | 6.47 (1.025)
  Leukocytes, Day 3 | 8.00 (4.384) | 5.30 (1.499)
  Leukocytes, Day 7 | 7.65 (3.606) | 5.58 (1.466)
  Leukocytes, Day 9 | 8.15 (5.020) | 5.75 (1.738)

14. Primary Outcome: Part 1: Absolute Values for Hematology Parameter: Erythrocytes
Description: Blood samples were collected at indicated time points to analyze erythrocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
10^12 cells per liter
  Baseline (Day -2) | 4.740 (0.0849) | 4.647 (0.3336)
  Day 3 | 5.010 (0.3253) | 4.820 (0.2626)
  Day 7 | 5.060 (0.3677) | 4.915 (0.3246)
  Day 9 | 5.065 (0.2475) | 4.852 (0.2556)

15. Primary Outcome: Part 1: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected at indicated time points to analyze hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Grams per liter
  Day 3 | 6.0 (5.66) | 5.5 (6.95)
  Day 7 | 8.0 (7.07) | 8.7 (8.29)
  Day 9 | 8.5 (2.12) | 5.8 (10.30)

16. Primary Outcome: Part 1: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected at indicated timepoints to analyze hemotocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Proportion of red blood cells in blood
  Day 3 | 0.0210 (0.02404) | 0.0128 (0.01779)
  Day 7 | 0.0250 (0.02404) | 0.0220 (0.02194)
  Day 9 | 0.0310 (0.01414) | 0.0142 (0.03330)

17. Primary Outcome: Part 1: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected at indicated time points to analyze erythrocytes mean corpuscular volume. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Femtoliter
  Day 3 | -0.40 (0.849) | -0.47 (0.403)
  Day 7 | -0.40 (0.283) | -0.37 (0.709)
  Day 9 | 0.50 (0.424) | -0.75 (0.802)

18. Primary Outcome: Part 1: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected at idicated time points to analyze erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Picograms
  Day 3 | -0.50 (0.141) | 0.08 (0.343)
  Day 7 | -0.35 (0.071) | 0.15 (0.501)
  Day 9 | -0.35 (0.354) | -0.02 (0.412)

19. Primary Outcome: Part 1: Change From Baseline in Hematology Parameter: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets and Leukocytes
Description: Blood samples were collected at indicated time points to analyze basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelets and leukocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
10^9 cells per liter
  Basophils, Day 3 | -0.005 (0.0212) | -0.003 (0.0137)
  Basophils, Day 7 | -0.005 (0.0212) | -0.008 (0.0160)
  Basophils, Day 9 | -0.010 (0.0424) | 0.008 (0.0098)
  Eosinophils, Day 3 | -0.025 (0.1909) | -0.022 (0.0462)
  Eosinophils, Day 7 | -0.030 (0.2828) | -0.035 (0.0497)
  Eosinophils, Day 9 | -0.045 (0.2616) | -0.040 (0.0559)
  Lymphocytes, Day 3 | 0.195 (0.2192) | -0.165 (0.2870)
  Lymphocytes, Day 7 | -0.005 (0.1626) | -0.153 (0.3222)
  Lymphocytes, Day 9 | -0.420 (0.3818) | 0.113 (0.2908)
  Monocytes, Day 3 | 0.020 (0.0566) | -0.075 (0.0885)
  Monocytes, Day 7 | -0.025 (0.0495) | -0.047 (0.1111)
  Monocytes, Day 9 | -0.060 (0.0566) | -0.028 (0.0755)
  Neutrophils, Day 3 | 0.290 (0.5233) | -0.895 (0.7988)
  Neutrophils, Day 7 | 0.195 (0.3182) | -0.632 (0.5515)
  Neutrophils, Day 9 | 1.205 (1.8455) | -0.742 (0.8588)
  Platelets, Day 3 | 5.0 (8.49) | -2.3 (17.68)
  Platelets, Day 7 | 15.5 (17.68) | 13.5 (29.49)
  Platelets, Day 9 | 11.0 (31.11) | 3.3 (36.74)
  Leukocytes, Day 3 | 0.65 (0.778) | -1.17 (0.942)
  Leukocytes, Day 7 | 0.30 (0.000) | -0.88 (0.818)
  Leukocytes, Day 9 | 0.80 (1.414) | -0.72 (1.011)

20. Primary Outcome: Part 1: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected at indicated time points to analyze the hematology parameter: Erythrocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
10^12 cells per liter
  Day 3 | 0.270 (0.2404) | 0.173 (0.2062)
  Day 7 | 0.320 (0.2828) | 0.268 (0.2513)
  Day 9 | 0.325 (0.1626) | 0.205 (0.3761)

21. Primary Outcome: Part 1: Absolute Values for Chemistry Parameters: Glucose, Cholesterol, Magnesium, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium, and Blood Urea Nitrogen
Description: Blood samples were collected at indicated time points to analyze glucose, cholesterol, magnesium, triglycerides, anion gap, calcium, carbon dioxide, chloride, phosphate, potassium, sodium, and blood urea nitrogen. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Millimoles per liter
  Glucose, Baseline (Day -2) | 5.050 (0.3960) | 4.682 (0.3788)
  Glucose, Day 3 | 4.495 (0.2333) | 4.745 (0.3566)
  Glucose, Day 7 | 4.465 (0.1202) | 4.728 (0.3251)
  Glucose, Day 9 | 4.635 (0.5162) | 4.605 (0.2660)
  Cholesterol, Baseline (Day-2) | 5.025 (0.6576) | 4.112 (0.6916)
  Cholesterol, Day 3 | 5.390 (1.1738) | 4.370 (0.5531)
  Cholesterol, Day 7 | 5.180 (1.1031) | 4.413 (0.7692)
  Cholesterol, Day 9 | 5.000 (0.9192) | 4.205 (0.8352)
  Magnesium, Baseline (Day -2) | 0.760 (0.0283) | 0.767 (0.0413)
  Magnesium, Day 3 | 0.800 (0.0849) | 0.787 (0.0301)
  Magnesium, Day 7 | 0.800 (0.0283) | 0.787 (0.0393)
  Magnesium, Day 9 | 0.800 (0.0283) | 0.813 (0.0301)
  Triglycerides, Baseline (Day -2) | 1.295 (0.8839) | 0.763 (0.2595)
  Triglycerides, Day 3 | 1.205 (0.1909) | 0.857 (0.2474)
  Triglycerides, Day 7 | 1.005 (0.2192) | 0.658 (0.2024)
  Triglycerides, Day 9 | 0.965 (0.1626) | 0.615 (0.1946)
  Anion gap, Baseline (Day-2) | 12.5 (0.71) | 10.3 (1.51)
  Anion gap, Day 3 | 11.5 (2.12) | 9.5 (1.52)
  Anion gap, Day 7 | 10.0 (0.00) | 10.3 (1.03)
  Anion gap, Day 9 | 11.0 (1.41) | 10.7 (1.75)
  Calcium, Baseline (Day -2) | 2.440 (0.0566) | 2.332 (0.0659)
  Calcium, Day 3 | 2.430 (0.0000) | 2.370 (0.0930)
  Calcium, Day 7 | 2.440 (0.0566) | 2.408 (0.1114)
  Calcium, Day 9 | 2.390 (0.0566) | 2.337 (0.0843)
  Carbon dioxide, Baseline (Day -2) | 29.0 (1.41) | 28.7 (1.75)
  Carbon dioxide, Day 3 | 30.0 (1.41) | 28.7 (2.16)
  Carbon dioxide, Day 7 | 30.5 (0.71) | 29.2 (1.60)
  Carbon dioxide, Day 9 | 30.0 (0.00) | 29.3 (2.25)
  Chloride, Baseline (Day -2) | 101.0 (2.83) | 103.7 (1.63)
  Chloride, Day 3 | 100.5 (2.12) | 102.7 (1.75)
  Chloride, Day 7 | 101.5 (0.71) | 102.2 (1.60)
  Chloride, Day 9 | 102.5 (0.71) | 103.2 (1.17)
  Phosphate, Baseline (Day -2) | 1.195 (0.0919) | 1.142 (0.1443)
  Phosphate, Day 3 | 1.210 (0.0707) | 1.238 (0.0519)
  Phosphate, Day 7 | 1.195 (0.0495) | 1.223 (0.1203)
  Phosphate, Day 9 | 1.130 (0.0000) | 1.212 (0.1983)
  Potassium, Baseline (Day -2) | 4.05 (0.071) | 4.10 (0.410)
  Potassium, Day 3 | 4.00 (0.141) | 4.28 (0.232)
  Potassium, Day 7 | 4.35 (0.071) | 4.22 (0.133)
  Potassium, Day 9 | 4.05 (0.071) | 4.20 (0.228)
  Sodium, Baseline (Day -2) | 138.5 (0.71) | 138.5 (1.64)
  Sodium, Day 3 | 138.0 (1.41) | 136.5 (1.05)
  Sodium, Day 7 | 138.0 (0.00) | 137.7 (1.51)
  Sodium, Day 9 | 139.5 (2.12) | 139.0 (0.89)
  Blood Urea Nitrogen, Baseline (Day -2) | 4.300 (1.4425) | 4.482 (1.2674)
  Blood Urea Nitrogen, Day 3 | 4.625 (1.2374) | 4.648 (0.6614)
  Blood Urea Nitrogen, Day 7 | 5.230 (0.7778) | 4.690 (0.6622)
  Blood Urea Nitrogen, Day 9 | 4.715 (0.4031) | 4.332 (0.7889)

22. Primary Outcome: Part 1: Absolute Values for Chemistry Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Gamma-glutamyl Transferase (GGT), Creatine Kinase, and Lactate Dehydrogenase
Description: Blood samples were collected at indicated time points to analyze ALT, ALP, AST, GGT, creatine kinase, and lactate dehydrogenase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
International units per liter
  ALT, Baseline (Day -2), | 33.0 (28.28) | 19.7 (10.97)
  ALT, Day 3 | 37.5 (33.23) | 16.8 (7.94)
  ALT, Day 7 | 33.5 (26.16) | 17.7 (5.92)
  ALT, Day 9 | 28.5 (23.33) | 18.2 (8.75)
  ALP, Baseline (Day -2) | 73.0 (22.63) | 54.3 (26.79)
  ALP, Day 3 | 76.5 (23.33) | 50.0 (15.05)
  ALP, Day 7 | 75.0 (26.87) | 54.8 (16.22)
  ALP, Day 9 | 75.5 (26.16) | 54.5 (17.44)
  AST, Baseline (Day -2) | 25.0 (9.90) | 19.8 (6.49)
  AST, Day 3 | 24.5 (12.02) | 17.5 (2.35)
  AST, Day 7 | 21.5 (7.78) | 18.0 (2.53)
  AST, Day 9 | 18.0 (5.66) | 17.5 (3.99)
  GGT, Baseline (Day -2) | 21.0 (14.14) | 11.0 (3.22)
  GGT, Day 3 | 21.5 (14.85) | 10.8 (3.37)
  GGT, Day 7 | 20.0 (14.14) | 12.0 (3.29)
  GGT, Day 9 | 19.5 (13.44) | 12.0 (3.69)
  Creatine kinase, Baseline (Day -2) | 93.0 (50.91) | 160.7 (124.55)
  Creatine kinase, Day 3 | 64.5 (24.75) | 91.2 (69.29)
  Creatine kinase, Day 7 | 71.5 (53.03) | 71.5 (53.73)
  Creatine kinase, Day 9 | 60.5 (34.65) | 75.5 (56.79)
  Lactate dehydrogenase, Baseline (Day -2) | 161.5 (36.06) | 132.0 (22.04)
  Lactate dehydrogenase, Day 3 | 150.0 (46.67) | 113.3 (22.55)
  Lactate dehydrogenase, Day 7 | 142.0 (22.63) | 115.8 (22.05)
  Lactate dehydrogenase, Day 9 | 133.0 (24.04) | 114.5 (26.10)

23. Primary Outcome: Part 1: Absolute Values for Chemistry Parameters: Creatinine, Urate, Total Bilirubin, and Direct Bilirubin
Description: Blood samples were collected at indicated timepoints to analyze creatinine, urate, total bilirubin, and direct bilirubin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 3, Day 7, Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Micromoles per liter
  Creatinine, Baseline (Day -2) | 89.75 (16.900) | 74.85 (15.104)
  Creatinine, Day 3 | 83.10 (13.718) | 72.20 (8.322)
  Creatinine, Day 7 | 86.60 (14.991) | 70.13 (8.411)
  Creatinine, Day 9 | 85.30 (10.607) | 71.00 (8.919)
  Urate, Baseline (Day -2) | 363.0 (0.00) | 274.5 (72.37)
  Urate, Day 3 | 351.0 (50.91) | 259.0 (61.48)
  Urate, Day 7 | 365.5 (54.45) | 246.0 (60.52)
  Urate, Day 9 | 348.0 (55.15) | 257.0 (59.67)
  Total Bilirubin, Baseline (Day -2) | 5.60 (1.697) | 7.00 (3.033)
  Total Bilirubin, Day 3 | 8.55 (0.212) | 9.63 (3.059)
  Total Bilirubin, Day 7 | 8.75 (0.212) | 11.33 (5.201)
  Total Bilirubin, Day 9 | 7.80 (1.556) | 10.20 (5.043)
  Direct Bilirubin, Baseline (Day -2) | 0.95 (0.354) | 1.42 (0.605)
  Direct Bilirubin, Day 3 | 1.45 (0.071) | 1.68 (0.571)
  Direct Bilirubin, Day 7 | 1.60 (0.141) | 2.10 (1.016)
  Direct Bilirubin, Day 9 | 1.55 (0.212) | 2.05 (0.862)

24. Primary Outcome: Part 1: Absolute Values for Chemistry Parameters: Albumin, Globulin, and Total Protein
Description: Blood samples were collected at indicated timepoints to analyze albumin, globulin, and total protein. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 3, Day 7, Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Grams per liter
  Albumin, Baseline (Day -2) | 46.5 (2.12) | 43.0 (3.03)
  Albumin, Day 3 | 46.0 (1.41) | 41.8 (3.31)
  Albumin, Day 7 | 47.5 (0.71) | 44.3 (3.61)
  Albumin, Day 9 | 45.5 (0.71) | 43.2 (2.64)
  Globulin, Baseline (Day -2) | 26.5 (2.12) | 25.5 (5.13)
  Globulin, Day 3 | 26.0 (0.00) | 27.7 (2.34)
  Globulin, Day 7 | 25.0 (1.41) | 27.8 (3.66)
  Globulin, Day 9 | 25.5 (0.71) | 27.5 (4.28)
  Total protein, Baseline (Day -2) | 73.0 (4.24) | 68.5 (5.47)
  Total protein, Day 3 | 72.0 (1.41) | 69.5 (3.27)
  Total protein, Day 7 | 72.5 (2.12) | 72.2 (4.07)
  Total Bilirubin, Day 9 | 71.0 (1.41) | 70.7 (4.76)

25. Primary Outcome: Part 1: Absolute Values for Chemistry Parameters: Amylase and Lipase
Description: Blood samples were collected at indicated timepoints to analyze amylase and lipase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Units per liter
  Amylase, Baseline (Day -2) | 64.5 (26.16) | 63.8 (22.54)
  Amylase, Day 3 | 64.0 (33.94) | 61.8 (25.31)
  Amylase, Day 7 | 67.0 (45.25) | 62.8 (22.45)
  Amylase, Day 9 | 64.5 (41.72) | 59.5 (22.05)
  Lipase, Baseline (Day -2) | 33.5 (20.51) | 35.5 (11.84)
  Lipase, Day 3 | 18.5 (2.12) | 30.2 (12.24)
  Lipase, Day 7 | 19.5 (3.54) | 32.3 (16.24)
  Lipase, Day 9 | 18.5 (3.54) | 29.3 (11.29)

26. Primary Outcome: Part 1: Change From Baseline in Chemistry Parameters: Glucose, Cholesterol, Magnesium, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium, Blood Urea Nitrogen
Description: Blood samples were collected at indicated time points to analyze glucose, cholesterol, magnesium, triglycerides, anion gap, calcium, carbon dioxide, chloride, phosphate, potassium, sodium, and blood urea nitrogen. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Millimoles per liter
  Glucose, Day 3 | -0.555 (0.6293) | 0.063 (0.3773)
  Glucose, Day 7 | -0.585 (0.5162) | 0.047 (0.2914)
  Glucose, Day 9 | -0.415 (0.9122) | -0.077 (0.3626)
  Cholesterol, Day 3 | 0.365 (0.5162) | 0.258 (0.3570)
  Cholesterol, Day 7 | 0.155 (0.4455) | 0.302 (0.2662)
  Cholesterol, Day 9 | -0.025 (0.2616) | 0.093 (0.2144)
  Magnesium, Day 3 | 0.040 (0.0566) | 0.020 (0.0335)
  Magnesium, Day 7 | 0.040 (0.0000) | 0.020 (0.0551)
  Magnesium, Day 9 | 0.040 (0.0000) | 0.047 (0.0468)
  Triglycerides, Day 3 | -0.090 (0.6930) | 0.093 (0.2432)
  Triglycerides, Day 7 | -0.290 (0.6647) | -0.105 (0.2076)
  Triglycerides, Day 9 | -0.330 (0.7212) | -0.148 (0.2494)
  Anion gap, Day 3 | -1.0 (1.41) | -0.8 (1.60)
  Anion gap, Day 7 | -2.5 (0.71) | 0.0 (1.90)
  Anion gap, Day 9 | -1.5 (2.12) | 0.3 (2.50)
  Calcium, Day 3 | -0.010 (0.0566) | 0.038 (0.0527)
  Calcium, Day 7 | 0.000 (0.1131) | 0.077 (0.0712)
  Calcium, Day 9 | -0.050 (0.1131) | 0.005 (0.0558)
  Carbon dioxide, Day 3 | 1.0 (2.83) | 0.0 (2.00)
  Carbon dioxide, Day 7 | 1.5 (0.71) | 0.5 (0.84)
  Carbon dioxide, Day 9 | 1.0 (1.41) | 0.7 (1.86)
  Chloride, Day 3 | -0.5 (0.71) | -1.0 (1.55)
  Chloride, Day 7 | 0.5 (2.12) | -1.5 (1.97)
  Chloride, Day 9 | 1.5 (2.12) | -0.5 (1.64)
  Phosphate, Day 3 | 0.015 (0.1626) | 0.097 (0.1136)
  Phosphate, Day 7 | 0.000 (0.1414) | 0.082 (0.1625)
  Phosphate, Day 9 | -0.065 (0.0919) | 0.070 (0.1898)
  Potassium, Day 3 | -0.05 (0.071) | 0.18 (0.366)
  Potassium, Day 7 | 0.30 (0.141) | 0.12 (0.331)
  Potassium, Day 9 | 0.00 (0.000) | 0.10 (0.363)
  Sodium, Day 3 | -0.5 (0.71) | -2.0 (1.90)
  Sodium, Day 7 | -0.5 (0.71) | -0.8 (2.04)
  Sodium, Day 9 | 1.0 (1.41) | 0.5 (1.87)
  Blood Urea Nitrogen, Day 3 | 0.325 (0.2051) | 0.167 (1.4356)
  Blood Urea Nitrogen, Day 7 | 0.930 (0.6647) | 0.208 (1.5113)
  Blood Urea Nitrogen, Day 9 | 0.415 (1.0394) | -0.150 (1.2510)

27. Primary Outcome: Part 1: Change From Baseline in Chemistry Parameters: ALT, ALP, AST, GGT, Creatine Kinase, Lactate Dehydrogenase
Description: Blood samples were collected at indicated time points to analyze ALT, ALP, AST, GGT, creatine kinase, and lactate dehydrogenase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
International units per liter
  ALT, Day 3 | 4.5 (4.95) | -2.8 (3.71)
  ALT, Day 7 | 0.5 (2.12) | -2.0 (9.70)
  ALT, Day 9 | -4.5 (4.95) | -1.5 (12.77)
  ALP, Day 3 | 3.5 (0.71) | -4.3 (12.14)
  ALP, Day 7 | 2.0 (4.24) | 0.5 (12.53)
  ALP, Day 9 | 2.5 (3.54) | 0.2 (10.80)
  AST, Day 3 | -0.5 (2.12) | -2.3 (5.50)
  AST, Day 7 | -3.5 (2.12) | -1.8 (7.91)
  AST, Day 9 | -7.0 (4.24) | -2.3 (8.80)
  GGT, Day 3 | 0.5 (0.71) | -0.2 (1.17)
  GGT, Day 7 | -1.0 (0.00) | 1.0 (0.89)
  GGT, Day 9 | -1.5 (0.71) | 1.0 (0.89)
  Creatine kinase, Day 3 | -28.5 (26.16) | -69.5 (104.08)
  Creatine kinase, Day 7 | -21.5 (2.12) | -89.2 (121.90)
  Creatine kinase, Day 9 | -32.5 (16.26) | -85.2 (127.35)
  Lactate dehydrogenase, Day 3 | -11.5 (10.61) | -18.7 (9.27)
  Lactate dehydrogenase, Day 7 | -19.5 (13.44) | -16.2 (9.99)
  Lactate dehydrogenase, Day 9 | -28.5 (12.02) | -17.5 (19.41)

28. Primary Outcome: Part 1: Change From Baseline in Chemistry Parameters: Creatinine, Urate, Total Bilirubin, Direct Bilirubin
Description: Blood samples were collected at indicated timepoints to analyze creatinine, urate, total bilirubin, and direct bilirubin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Micromoles per liter
  Creatinine, Day 3 | -6.65 (3.182) | -2.65 (12.451)
  Creatinine, Day 7 | -3.15 (1.909) | -4.72 (10.794)
  Creatinine, Day 9 | -4.45 (6.293) | -3.85 (10.095)
  Urate, Day 3 | -12.0 (50.91) | -15.5 (33.59)
  Urate, Day 7 | 2.5 (54.45) | -28.5 (32.72)
  Urate, Day 9 | -15.0 (55.15) | -17.5 (23.86)
  Total Bilirubin, Day 3 | 2.95 (1.909) | 2.63 (2.534)
  Total Bilirubin, Day 7 | 3.15 (1.485) | 4.33 (2.653)
  Total Bilirubin, Day 9 | 2.20 (0.141) | 3.20 (2.225)
  Direct Bilirubin, Day 3 | 0.50 (0.283) | 0.27 (0.535)
  Direct Bilirubin, Day 7 | 0.65 (0.212) | 0.68 (0.534)
  Direct Bilirubin, Day 9 | 0.60 (0.141) | 0.63 (0.398)

29. Primary Outcome: Part 1: Change From Baseline in Chemistry Parameters: Albumin, Globulin, and Total Protein
Description: Blood samples were collected at indicated timepoints to analyze albumin, globulin, and total protein. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Grams per liter
  Albumin, Day 3 | -0.5 (3.54) | -1.2 (0.75)
  Albumin, Day 7 | 1.0 (2.83) | 1.3 (2.94)
  Albumin, Day 9 | -1.0 (2.83) | 0.2 (2.14)
  Globulin, Day 3 | -0.5 (2.12) | 2.2 (3.49)
  Globulin, Day 7 | -1.5 (3.54) | 2.3 (2.07)
  Globulin, Day 9 | -1.0 (2.83) | 2.0 (1.41)
  Total protein, Day 3 | -1.0 (5.66) | 1.0 (4.20)
  Total protein, Day 7 | -0.5 (6.36) | 3.7 (4.80)
  Total Bilirubin, Day 9 | -2.0 (5.66) | 2.2 (3.19)

30. Primary Outcome: Part 1: Change From Baseline in Chemistry Parameters: Amylase and Lipase
Description: Blood samples were collected at indicated timepoints to analyze amylase and lipase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Units per liter
  Amylase, Day 3 | -0.5 (7.78) | -2.0 (8.72)
  Amylase, Day 7 | 2.5 (19.09) | -1.0 (3.95)
  Amylase, Day 9 | 0.0 (15.56) | -4.3 (5.57)
  Lipase, Day 3 | -15.0 (18.38) | -5.3 (8.12)
  Lipase, Day 7 | -14.0 (16.97) | -3.2 (7.73)
  Lipase, Day 9 | -15.0 (16.97) | -6.2 (4.31)

31. Primary Outcome: Part 1: Absolute Values for Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected at indicated time points to analyze the urine specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Ratio
  Baseline (Day -2) | 1.0080 (0.00707) | 1.0092 (0.00574)
  Day 3 | 1.0150 (0.00141) | 1.0125 (0.00565)
  Day 7 | 1.0190 (0.00283) | 1.0167 (0.00450)
  Day 9 | 1.0145 (0.00212) | 1.0097 (0.00557)

32. Primary Outcome: Part 1: Absolute Values for Urinalysis Parameter: Potential of Hydrogen (pH)
Description: Urine samples were collected at indicated time points to analyze the urine pH by dipstick test. The dipstick test gives results in a semi-quantitative manner indicating proportional concentrations in the urine sample. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
pH
  Baseline (Day -2) | 6.50 (0.707) | 7.08 (0.585)
  Day 3 | 6.50 (0.707) | 6.33 (0.606)
  Day 7 | 6.25 (0.354) | 6.25 (0.524)
  Day 9 | 6.50 (0.707) | 6.25 (0.418)

33. Primary Outcome: Part 1: Change From Baseline in Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected at indicated time points to analyze the urine specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Ratio
  Day 3 | 0.0070 (0.00566) | 0.0033 (0.00653)
  Day 7 | 0.0110 (0.00424) | 0.0075 (0.00731)
  Day 9 | 0.0065 (0.00495) | 0.0005 (0.00912)

34. Primary Outcome: Part 1: Change From Baseline in Urinalysis Parameter: pH
Description: Urine samples were collected at indicated time points to analyze the urine pH by dipstick test. The dipstick test gives results in a semi-quantitative manner indicating proportional concentrations in the urine sample. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 3, Day 7, and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
pH
  Day 3 | 0.00 (1.414) | -0.75 (0.612)
  Day 7 | -0.25 (1.061) | -0.83 (0.408)
  Day 9 | 0.00 (1.414) | -0.83 (0.258)

35. Primary Outcome: Part 1: Number of Participants With Clinically Significant Abnormal 12-Lead Electrocardiogram (ECG) Findings
Description: A 12-lead ECG was recorded with the participant in a supine position. 12-lead ECGs were obtained by using an automated ECG machine. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for number of participants with clinically significant abnormal 12-Lead ECG findings has reported
Time Frame: Baseline(Day-2), Day1: 2 Hours, 4 Hours, 6 Hours; Day 4: 2 Hours, 4 Hours, 6 Hours, Day 7: 2 Hours, 4 Hours, 6 Hours and Day 9
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Participants
  Baseline (Day -2) | 0 | 0
  Day 1: 2 hours | 0 | 0
  Day 1: 4 hours | 0 | 0
  Day 1: 6 hours | 0 | 0
  Day 4: 2 hours | 0 | 0
  Day 4: 4 hours | 0 | 0
  Day 4: 6 hours | 0 | 0
  Day 7: 2 hours | 0 | 0
  Day 7: 4 hours | 0 | 0
  Day 7: 6 hours | 0 | 0
  Day 9 | 0 | 0

36. Primary Outcome: Part 1: Absolute Values for Vital Parameters: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in the semi-recumbent or supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Pre-dose, Day 1), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8 and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters (mm) of mercury
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Millimeters (mm) of mercury
  SBP, Baseline (Pre-dose, Day 1) | 120.0 (1.41) | 109.2 (12.22)
  SBP, Day 2 | 115.5 (0.71) | 103.8 (10.42)
  SBP, Day 3 | 123.0 (2.83) | 106.8 (9.87)
  SBP, Day 4 | 121.5 (17.68) | 107.5 (13.74)
  SBP, Day 5 | 111.5 (9.19) | 105.3 (5.20)
  SBP, Day 6 | 114.0 (15.56) | 107.0 (6.57)
  SBP, Day 7 | 117.5 (4.95) | 107.7 (10.07)
  SBP, Day 8 | 125.0 (1.41) | 109.0 (6.48)
  SBP, Day 9 | 127.0 (5.66) | 109.8 (7.81)
  DBP, Baseline (Pre-dose, Day 1) | 74.0 (4.24) | 61.5 (8.22)
  DBP, Day 2 | 70.5 (4.95) | 59.8 (5.74)
  DBP, Day 3 | 76.0 (5.66) | 59.7 (3.14)
  DBP, Day 4 | 66.0 (14.14) | 64.0 (9.90)
  DBP, Day 5 | 69.5 (21.92) | 62.3 (5.57)
  DBP, Day 6 | 65.5 (12.02) | 61.2 (4.49)
  DBP, Day 7 | 72.0 (11.31) | 63.7 (5.79)
  DBP, Day 8 | 67.0 (8.49) | 64.5 (9.65)
  DBP, Day 9 | 69.5 (9.19) | 64.7 (7.50)

37. Primary Outcome: Part 1: Absolute Values for Vital Parameter: Pulse Rate
Description: Pulse rate was measured in the semi-recumbent or supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Pre-dose, Day 1), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8 and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Beats per minute (bpm)
  Baseline (Pre-dose, Day 1 ) | 70.5 (7.78) | 67.8 (13.44)
  Day 2 | 63.0 (7.07) | 68.7 (10.60)
  Day 3 | 70.5 (2.12) | 65.0 (10.24)
  Day 4 | 71.0 (5.66) | 68.8 (12.29)
  Day 5 | 67.0 (14.14) | 72.5 (12.32)
  Day 6 | 66.5 (3.54) | 67.2 (8.57)
  Day 7 | 70.0 (7.07) | 70.5 (7.50)
  Day 8 | 70.0 (8.49) | 81.3 (9.63)
  Day 9 | 73.0 (2.83) | 67.8 (9.02)

38. Primary Outcome: Part 1: Absolute Values for Vital Parameter: Temperature
Description: Temperature was measured in the semi-recumbent or supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions.Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Pre-dose, Day 1), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8 and Day 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part 1 : Placebo | Part 1 : GSK3640254 500 mg
Number analyzed (Participants) | 2 | 6
Degrees Celsius
  Baseline (Pre-dose, Day 1) | 35.90 (0.424) | 36.50 (0.341)
  Day 2 | 36.10 (0.424) | 36.53 (0.225)
  Day 3 | 36.10 (0.283) | 36.58 (0.264)
  Day 4 | 36.15 (0.354) | 36.52 (0.479)
  Day 5 | 36.35 (0.354) | 36.58 (0.360)
  Day 6 | 36.45 (0.354) | 36.47 (0.250)
  Day 7 | 35.95 (0.495) | 36.47 (0.383)
  Day 8 | 36.35 (0.071) | 36.63 (0.280)
  Day 9 | 36.35 (0.212) | 36.47 (0.234)

39. Primary Outcome: Part 2: Placebo-corrected Change From Baseline in QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF) Following Administration of GSK3640254 100 mg and GSK3640254 500 mg Using Concentration-QTc (C-QTc) Analysis
Description: Twelve-lead ECGs were recorded in participant using automated ECG machine & performed with participant in supine position after a rest of at least 10 minutes.Baseline was defined as the latest pre-dose assessment with a non-missing value for each visit. Change from Baseline was calculated by subtracting Baseline value from post dose value. Placebo-corrected change from Baseline in QT interval corrected for heart rate using Fridericia's formula (QTcF) was calculated as difference in model-predicted mean change from Baseline in QTcF between treatment groups using C-QTc analysis. A linear mixed-effects model with change from Baseline in QTcF as the dependent variable, time-matched GSK3640254 plasma concentration as a fixed effect, centered Baseline as additional covariate,treatment &time as categorical factors, & a random intercept & slope per participant. In all calculations, concentrations in participants who received placebo were set to 0.
Time Frame: Baseline (Pre-dose, Day 1) and up to Day 7
Population: PK/QTc Population comprised of all participants who are in both QT/QTc and PK concentration Populations with at least 1 pair of post-dose PK and change from Baseline in QTc data from the same time point as well as participants in the QT/QTc Population who received placebo. Only those participants with data available at specified time points were analyzed. This outcome measure(OM) intended to provide Placebo-corrected data. Summary of change from Baseline data is provided in OM43.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Milliseconds (ms)
Groups:
- Part 2: GSK3640254 100 mg: Participants received therapeutic dose of GSK3640254 100 mg once daily from Days 1 through 7 in each Treatment Period of Part 2 of the study.
- Part 2: GSK3640254 500 mg: Participants received supratherapeutic dose of GSK3640254 500 mg once daily from Days 1 through 7 in each Treatment Period of Part 2 of the study.
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 40 | 39
Milliseconds (ms) | 2.72 [2.04 to 3.39] | 11.49 [9.24 to 13.73]

40. Primary Outcome: Part 2: Plasma Concentration of GSK3640254
Description: Blood samples were collected at indicated time points to analyze the plasma concentration of GSK3640254.
Time Frame: Pre-dose and 30 minutes, 1 Hour, 2 Hour, 3 Hours, 3 Hours 30 minutes, 4 Hours, 4 Hours 30 minutes, 5 Hours, 6 Hours, 8 Hours, 10 Hours, 12 Hours, 24 Hours post-dose on Day 7 in each treatment period
Population: Pharmacokinetic Concentration Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 40 | 40
Nanograms per milliliter
  Pre-dose, Day 7 | 496.0 (209.03) | 2357 (1137.1)
  30 minutes, Day 7 | 462.3 (188.61) | 2252 (1266.0)
  1 Hour, Day 7 | 486.6 (198.56) | 2339 (1289.3)
  2 Hour, Day 7 | 587.8 (298.21) | 2779 (1670.6)
  3 Hour, Day 7 | 682.4 (329.52) | 3372 (1757.9)
  3 Hours 30 minutes, Day 7 | 738.6 (368.38) | 3698 (1812.2)
  4 Hour, Day 7 | 765.5 (349.05) | 4011 (1880.5)
  4 Hours 30 minutes, Day 7 | 782.4 (318.09) | 4157 (1927.0)
  5 Hour, Day 7 | 811.3 (326.24) | 4172 (1804.9)
  6 Hour, Day 7 | 769.8 (265.82) | 4102 (1719.5)
  8 Hour, Day 7 | 740.9 (280.65) | 3762 (1727.0)
  10 Hour, Day 7 | 698.7 (280.28) | 3564 (1603.7)
  12 Hour, Day 7 | 625.4 (231.50) | 3098 (1347.5)
  24 Hour, Day 7 | 469.9 (183.24) | 2257 (1127.6)

41. Primary Outcome: Part 2: Plasma Concentration of Major Metabolites of GSK3640254
Description: as for outcome 7
Time Frame: as for outcome 40
Population: as for outcome 7
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 0 | 0

42. Secondary Outcome: Part 2: Change From Baseline in Heart Rate (HR) - For GSK3640254 100 mg, GSK3640254 500 mg and Placebo Arms
Description: Twelve-lead ECGs were recorded in participant using an automated ECG machine. Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Pre-dose, Day 1), Day 7 : Predose and 0.5, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 Hours post dose
Population: QT/QTc Population comprised of all participants in the safety population with measurements at baseline as well as on-treatment with at least 1 post-dose time point with a valid change from Baseline in QTc value. Only those participants with data available at specified time points were analyzed.
Measure: Least Squares Mean (90% Confidence Interval); unit: Beats per minute
Groups:
- Part 2: Placebo: Participants received placebo matching GSK3640254 from Days 1 through 7 in each Treatment Period of Part 2 of the study.
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg | Part 2: Placebo
Number analyzed (Participants) | 40 | 39 | 40
Beats per minute
  Day 7, Predose: number analyzed (Participants) | 40 | 37 | 38
  Day 7, Predose | 0.0 [-1.71 to 1.75] | 2.8 [1.03 to 4.56] | 0.3 [-1.42 to 2.08]
  Day7, 0.5 Hour Post-dose: number analyzed (Participants) | 39 | 38 | 40
  Day7, 0.5 Hour Post-dose | 4.4 [2.62 to 6.15] | 8.5 [6.71 to 10.27] | 4.6 [2.87 to 6.39]
  Day 7, 1 Hour Post-dose: number analyzed (Participants) | 39 | 37 | 40
  Day 7, 1 Hour Post-dose | 5.4 [3.70 to 7.06] | 9.1 [7.44 to 10.85] | 5.2 [3.51 to 6.86]
  Day7, 2 Hour Post-dose: number analyzed (Participants) | 40 | 37 | 40
  Day7, 2 Hour Post-dose | 5.9 [4.36 to 7.35] | 7.0 [5.47 to 8.51] | 4.5 [3.01 to 5.99]
  Day 7, 3 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 40
  Day 7, 3 Hour Post-dose | 4.1 [2.44 to 5.76] | 5.6 [3.88 to 7.24] | 2.7 [1.01 to 4.32]
  Day7, 3.5 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 38
  Day7, 3.5 Hour Post-dose | 4.5 [2.86 to 6.15] | 6.0 [4.29 to 7.63] | 2.8 [1.15 to 4.47]
  Day7, 4 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 39
  Day7, 4 Hour Post-dose | 3.7 [2.00 to 5.35] | 5.9 [4.22 to 7.62] | 2.6 [0.91 to 4.27]
  Day7, 4.5 Hour Post-dose: number analyzed (Participants) | 40 | 37 | 39
  Day7, 4.5 Hour Post-dose | 5.4 [3.43 to 7.41] | 6.9 [4.81 to 8.89] | 3.7 [1.65 to 5.66]
  Day7, 5 Hour Post-dose: number analyzed (Participants) | 39 | 36 | 38
  Day7, 5 Hour Post-dose | 5.0 [3.38 to 6.68] | 7.5 [5.82 to 9.18] | 3.4 [1.77 to 5.08]
  Day7, 6 Hour Post-dose: number analyzed (Participants) | 39 | 37 | 38
  Day7, 6 Hour Post-dose | 9.6 [7.68 to 11.58] | 12.7 [10.73 to 14.69] | 8.6 [6.64 to 10.56]
  Day7, 8 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 37
  Day7, 8 Hour Post-dose | 7.3 [5.56 to 9.11] | 10.5 [8.69 to 12.29] | 6.3 [4.46 to 8.06]
  Day7, 10 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 38
  Day7, 10 Hour Post-dose | 2.6 [0.93 to 4.31] | 7.0 [5.28 to 8.71] | 1.9 [0.16 to 3.57]
  Day7, 12 Hour Post-dose: number analyzed (Participants) | 40 | 39 | 37
  Day7, 12 Hour Post-dose | 8.5 [6.74 to 10.31] | 9.2 [7.38 to 10.98] | 8.1 [6.27 to 9.90]
  Day7, 24 Hour Post-dose: number analyzed (Participants) | 39 | 36 | 38
  Day7, 24 Hour Post-dose | 2.0 [0.29 to 3.80] | 3.3 [1.53 to 5.10] | -0.6 [-2.33 to 1.20]

43. Secondary Outcome: Part 2: Change From Baseline in QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF) - For GSK3640254 100 mg, GSK3640254 500 mg and Placebo Arms
Description: Twelve-lead ECGs were recorded in participant using automated ECG machine & performed with participant in supine position after a rest of at least 10 minutes.Baseline was defined as the latest pre-dose assessment with a non-missing value for each visit. Change from Baseline in QT interval corrected for heart rate using Fridericia's formula (QTcF) was calculated by subtracting Baseline value from post dose value.
Time Frame: Baseline (Pre-dose, Day 1), Day 7: Predose and 0.5, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 Hours post dose
Population: QT/QTc Population. Only those participants with data available at specified time points were analyzed.
Measure: Least Squares Mean (90% Confidence Interval); unit: Milliseconds
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg | Part 2: Placebo
Number analyzed (Participants) | 40 | 39 | 40
Milliseconds
  Day 7, Predose: number analyzed (Participants) | 40 | 37 | 38
  Day 7, Predose | 4.2 [2.47 to 5.88] | 9.8 [8.08 to 11.59] | 2.7 [1.01 to 4.46]
  Day7, 0.5 Hour Post-dose: number analyzed (Participants) | 39 | 38 | 40
  Day7, 0.5 Hour Post-dose | -0.9 [-2.76 to 1.03] | 5.3 [3.42 to 7.28] | -1.9 [-3.75 to 0.02]
  Day 7, 1 Hour Post-dose: number analyzed (Participants) | 39 | 37 | 40
  Day 7, 1 Hour Post-dose | 0.4 [-1.59 to 2.32] | 3.8 [1.79 to 5.80] | -0.3 [-2.22 to 1.68]
  Day7, 2 Hour Post-dose: number analyzed (Participants) | 40 | 37 | 40
  Day7, 2 Hour Post-dose | -2.2 [-4.36 to -0.03] | 2.6 [0.35 to 4.80] | -3.9 [-6.09 to -1.76]
  Day 7, 3 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 40
  Day 7, 3 Hour Post-dose | -2.8 [-4.95 to -0.65] | 3.7 [1.55 to 5.95] | -4.3 [-6.48 to -2.18]
  Day7, 3.5 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 38
  Day7, 3.5 Hour Post-dose | -2.9 [-4.89 to -0.97] | 4.8 [2.82 to 6.84] | -4.4 [-6.33 to -2.38]
  Day7, 4 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 39
  Day7, 4 Hour Post-dose | -2.0 [-3.90 to -0.17] | 5.6 [3.71 to 7.52] | -3.0 [-4.88 to -1.14]
  Day7, 4.5 Hour Post-dose: number analyzed (Participants) | 40 | 37 | 39
  Day7, 4.5 Hour Post-dose | -1.5 [-3.51 to 0.50] | 8.0 [5.95 to 10.08] | -2.6 [-4.57 to -0.53]
  Day7, 5 Hour Post-dose: number analyzed (Participants) | 39 | 36 | 38
  Day7, 5 Hour Post-dose | -1.1 [-3.00 to 0.81] | 8.3 [6.35 to 10.26] | -1.3 [-3.19 to 0.64]
  Day7, 6 Hour Post-dose: number analyzed (Participants) | 39 | 37 | 38
  Day7, 6 Hour Post-dose | -1.2 [-3.54 to 1.16] | 5.7 [3.30 to 8.10] | -2.9 [-5.25 to -0.52]
  Day7, 8 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 37
  Day7, 8 Hour Post-dose | -8.5 [-10.45 to -6.55] | 0.4 [-1.58 to 2.41] | -7.7 [-9.67 to -5.70]
  Day7, 10 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 38
  Day7, 10 Hour Post-dose | -4.0 [-5.84 to -2.26] | 4.4 [2.59 to 6.26] | -4.2 [-6.05 to -2.40]
  Day7, 12 Hour Post-dose: number analyzed (Participants) | 40 | 39 | 37
  Day7, 12 Hour Post-dose | -1.5 [-3.61 to 0.51] | 4.0 [1.88 to 6.06] | -2.0 [-4.12 to 0.10]
  Day7, 24 Hour Post-dose: number analyzed (Participants) | 39 | 36 | 38
  Day7, 24 Hour Post-dose | -0.5 [-2.50 to 1.42] | 7.1 [5.07 to 9.14] | -0.6 [-2.57 to 1.39]

44. Secondary Outcome: Part 2: Change From Baseline in PR Interval - For GSK3640254 100 mg, GSK3640254 500 mg and Placebo Arms
Description: Twelve-lead ECGs were recorded in participant using an automated ECG machine. Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Pre-dose, Day 1), Day 7: Predose and 0.5, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 Hours post dose
Population: QT/QTc Population. Only those participants with data available at specified time points were analyzed.
Measure: Least Squares Mean (90% Confidence Interval); unit: Milliseconds
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg | Part 2: Placebo
Number analyzed (Participants) | 40 | 39 | 40
Milliseconds
  Day 7, Predose: number analyzed (Participants) | 40 | 37 | 38
  Day 7, Predose | 2.5 [-1.09 to 6.10] | 3.1 [-0.51 to 6.74] | 1.1 [-2.56 to 4.66]
  Day7, 0.5 Hour Post-dose: number analyzed (Participants) | 39 | 38 | 40
  Day7, 0.5 Hour Post-dose | 3.6 [-0.05 to 7.23] | 5.7 [2.03 to 9.34] | 3.2 [-0.42 to 6.84]
  Day 7, 1 Hour Post-dose: number analyzed (Participants) | 39 | 37 | 40
  Day 7, 1 Hour Post-dose | 0.7 [-2.82 to 4.31] | -0.3 [-3.86 to 3.30] | -0.4 [-3.97 to 3.14]
  Day7, 2 Hour Post-dose: number analyzed (Participants) | 40 | 37 | 40
  Day7, 2 Hour Post-dose | -3.6 [-6.97 to -0.15] | -1.2 [-4.64 to 2.22] | -2.8 [-6.17 to 0.65]
  Day 7, 3 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 40
  Day 7, 3 Hour Post-dose | -4.3 [-7.79 to -0.76] | -2.6 [-6.18 to 0.89] | -4.7 [-8.20 to -1.16]
  Day7, 3.5 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 38
  Day7, 3.5 Hour Post-dose | -3.9 [-7.36 to -0.35] | -1.5 [-5.04 to 2.01] | -4.7 [-8.24 to -1.21]
  Day7, 4 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 39
  Day7, 4 Hour Post-dose | -3.4 [-6.82 to 0.05] | -2.9 [-6.38 to 0.53] | -4.6 [-8.06 to -1.17]
  Day7, 4.5 Hour Post-dose: number analyzed (Participants) | 40 | 37 | 39
  Day7, 4.5 Hour Post-dose | -4.7 [-8.21 to -1.16] | -4.3 [-7.82 to -0.72] | -5.3 [-8.88 to -1.81]
  Day7, 5 Hour Post-dose: number analyzed (Participants) | 39 | 36 | 38
  Day7, 5 Hour Post-dose | -3.9 [-7.36 to -0.44] | -3.7 [-7.15 to -0.18] | -3.9 [-7.41 to -0.47]
  Day7, 6 Hour Post-dose: number analyzed (Participants) | 39 | 37 | 38
  Day7, 6 Hour Post-dose | -3.8 [-7.37 to -0.27] | -3.9 [-7.43 to 0.29] | -4.1 [-7.61 to -0.50]
  Day7, 8 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 37
  Day7, 8 Hour Post-dose | -5.6 [-9.06 to -2.11] | -4.1 [-7.61 to -0.62] | -5.3 [-8.76 to -1.76]
  Day7, 10 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 38
  Day7, 10 Hour Post-dose | -3.9 [-7.36 to -0.49] | -3.9 [-7.35 to -0.46] | -5.0 [-8.44 to -1.55]
  Day7, 12 Hour Post-dose: number analyzed (Participants) | 40 | 39 | 37
  Day7, 12 Hour Post-dose | -3.0 [-6.46 to 0.39] | -1.8 [-5.23 to 1.63] | -3.6 [-7.05 to -0.17]
  Day7, 24 Hour Post-dose: number analyzed (Participants) | 39 | 36 | 38
  Day7, 24 Hour Post-dose | -0.5 [-3.99 to 2.92] | -0.9 [-4.40 to 2.57] | 0.9 [-2.56 to 4.38]

45. Secondary Outcome: Part 2: Change From Baseline in QRS Interval - For GSK3640254 100 mg, GSK3640254 500 mg and Placebo Arms
Description: as for outcome 42
Time Frame: Baseline (Pre-dose, Day 1), Day 7 : Predose and 0.5, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 Hours post dose
Population: QT/QTc Population. Only those participants with data available at specified time points were analyzed.
Measure: Least Squares Mean (90% Confidence Interval); unit: Milliseconds
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg | Part 2: Placebo
Number analyzed (Participants) | 40 | 39 | 40
Milliseconds
  Day 7, Predose: number analyzed (Participants) | 40 | 37 | 38
  Day 7, Predose | 0.5 [-0.07 to 1.00] | 1.0 [0.44 to 1.54] | 0.4 [-0.16 to 0.92]
  Day7, 0.5 Hour Post-dose: number analyzed (Participants) | 39 | 38 | 40
  Day7, 0.5 Hour Post-dose | 0.7 [0.19 to 1.27] | 1.1 [0.52 to 1.62] | 0.5 [-0.02 to 1.06]
  Day 7, 1 Hour Post-dose: number analyzed (Participants) | 39 | 37 | 40
  Day 7, 1 Hour Post-dose | 0.5 [-0.05 to 0.98] | 0.8 [0.28 to 1.33] | 0.1 [-0.40 to 0.64]
  Day7, 2 Hour Post-dose: number analyzed (Participants) | 40 | 37 | 40
  Day7, 2 Hour Post-dose | 0.4 [-0.17 to 0.88] | 0.6 [0.05 to 1.12] | -0.1 [-0.64 to 0.41]
  Day 7, 3 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 40
  Day 7, 3 Hour Post-dose | 0.6 [0.11 to 1.14] | 0.5 [-0.01 to 1.04] | 0.1 [-0.42 to 0.61]
  Day7, 3.5 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 38
  Day7, 3.5 Hour Post-dose | 0.6 [0.07 to 1.20] | 0.9 [0.34 to 1.48] | 0.3 [-0.27 to 0.86]
  Day7, 4 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 39
  Day7, 4 Hour Post-dose | 0.9 [0.38 to 1.49] | 1.1 [0.57 to 1.70] | 0.6 [0.07 to 1.18]
  Day7, 4.5 Hour Post-dose: number analyzed (Participants) | 40 | 37 | 39
  Day7, 4.5 Hour Post-dose | 1.1 [0.51 to 1.63] | 1.3 [0.69 to 1.84] | 0.9 [0.32 to 1.44]
  Day7, 5 Hour Post-dose: number analyzed (Participants) | 39 | 36 | 38
  Day7, 5 Hour Post-dose | 1.3 [0.66 to 1.85] | 1.5 [0.85 to 2.07] | 1.0 [0.42 to 1.62]
  Day7, 6 Hour Post-dose: number analyzed (Participants) | 39 | 37 | 38
  Day7, 6 Hour Post-dose | 1.3 [0.62 to 1.97] | 1.3 [0.66 to 2.02] | 1.2 [0.51 to 1.85]
  Day7, 8 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 37
  Day7, 8 Hour Post-dose | 0.5 [-0.14 to 1.14] | 0.9 [0.24 to 1.54] | 0.2 [-0.43 to 0.86]
  Day7, 10 Hour Post-dose: number analyzed (Participants) | 40 | 38 | 38
  Day7, 10 Hour Post-dose | 1.1 [0.48 to 1.66] | 1.2 [0.61 to 1.82] | 0.6 [-0.01 to 1.19]
  Day7, 12 Hour Post-dose: number analyzed (Participants) | 40 | 39 | 37
  Day7, 12 Hour Post-dose | 0.8 [0.20 to 1.39] | 0.7 [0.09 to 1.29] | 0.2 [-0.36 to 0.83]
  Day7, 24 Hour Post-dose: number analyzed (Participants) | 39 | 36 | 38
  Day7, 24 Hour Post-dose | 0.4 [-0.26 to 1.06] | 0.9 [0.22 to 1.58] | -0.5 [-1.13 to 0.20]

46. Secondary Outcome: Part 2: Placebo-corrected Change From Baseline in QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF) Following Administration of GSK3640254 100 mg and GSK3640254 500 mg By-time Point Analysis
Description: Twelve-lead ECGs were recorded in participant using automated ECG machine & performed with participant in supine position after a rest of at least 10 minutes.Baseline was defined as the latest pre-dose assessment with a non-missing value for each visit. Change from Baseline was calculated by subtracting Baseline value from post dose value. Placebo-corrected change from Baseline in QT interval corrected for heart rate using Fridericia's formula (QTcF) was calculated as model-predicted mean change from Baseline in QTcF in GSK3640254 group minus model-predicted mean change from Baseline in QTcF in the placebo group (by-time point analysis). Time point analysis was performed based on a linear mixed-effects model: Change from Baseline in QTcF = Time + Treatment + Time*Treatment +Baseline QTcF + Period + Sequence. An unstructured covariance structure was used to specify the repeated measures (time within participant and period). A random intercept per participant was also included.
Time Frame: Baseline (Pre-dose, Day 1), Day 7 : Predose and 0.5, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 Hours post dose
Population: QT/QTc Population. Only those participants with data available at specified time points were analyzed. This outcome measure is intended to provide Placebo-corrected data. Placebo and treatment wise change from Baseline data is provided in outcome measure number 43.
Measure: Least Squares Mean (90% Confidence Interval); unit: Milliseconds
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 40 | 39
Milliseconds
  Day7, Predose: number analyzed (Participants) | 40 | 37
  Day7, Predose | 1.4 [-0.88 to 3.77] | 7.1 [4.74 to 9.46]
  Day7, 0.5 Hour Post-dose: number analyzed (Participants) | 39 | 38
  Day7, 0.5 Hour Post-dose | 1.0 [-1.60 to 3.59] | 7.2 [4.59 to 9.83]
  Day7, 1 Hour Post-dose: number analyzed (Participants) | 39 | 37
  Day7, 1 Hour Post-dose | 0.6 [-2.06 to 3.33] | 4.1 [1.34 to 6.79]
  Day7, 2 Hour Post-dose: number analyzed (Participants) | 40 | 37
  Day7, 2 Hour Post-dose | 1.7 [-1.27 to 4.73] | 6.5 [3.46 to 9.55]
  Day7, 3 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 3 Hour Post-dose | 1.5 [-1.45 to 4.51] | 8.1 [5.06 to 11.09]
  Day7, 3.5 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 3.5 Hour Post-dose | 1.4 [-1.30 to 4.13] | 9.2 [6.44 to 11.93]
  Day7, 4 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 4 Hour Post-dose | 1.0 [-1.59 to 3.54] | 8.6 [6.03 to 11.22]
  Day7, 4.5 Hour Post-dose: number analyzed (Participants) | 40 | 37
  Day7, 4.5 Hour Post-dose | 1.0 [-1.73 to 3.82] | 10.6 [7.75 to 13.38]
  Day7, 5 Hour Post-dose: number analyzed (Participants) | 39 | 36
  Day7, 5 Hour Post-dose | 0.2 [-2.44 to 2.80] | 9.6 [6.92 to 12.24]
  Day7, 6 Hour Post-dose: number analyzed (Participants) | 39 | 37
  Day7, 6 Hour Post-dose | 1.7 [-1.58 to 4.97] | 8.6 [5.27 to 11.89]
  Day7, 8 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 8 Hour Post-dose | -0.8 [-3.54 to 1.90] | 8.1 [5.34 to 10.85]
  Day7, 10 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 10 Hour Post-dose | 0.2 [-2.30 to 2.65] | 8.6 [6.14 to 11.15]
  Day7, 12 Hour Post-dose | 0.5 [-2.43 to 3.35] | 6.0 [3.07 to 8.89]
  Day7, 24 Hour Post-dose: number analyzed (Participants) | 39 | 36
  Day7, 24 Hour Post-dose | 0.1 [-2.66 to 2.76] | 7.7 [4.94 to 10.45]

47. Secondary Outcome: Part 2: Placebo-corrected Change From Baseline in HR Following Administration of GSK3640254 100 mg and GSK3640254 500 mg
Description: Twelve-lead ECGs were recorded in participant using an automated ECG machine. Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Baseline is defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value. Placebo-corrected change from Baseline in HR was calculated as model-predicted mean change from Baseline in HR in GSK3640254 group minus model-predicted mean change from Baseline in HR in the placebo group.
Time Frame: Baseline (Pre-dose, Day 1) Day 7: Predose and 0.5, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 Hours post dose
Population: QT/QTc Population. Only those participants with data available at specified time points were analyzed. This outcome measure is intended to provide Placebo-corrected data. Placebo and treatment wise change from Baseline data is provided in outcome measure number 42.
Measure: Least Squares Mean (90% Confidence Interval); unit: Beats per minute
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 40 | 39
Beats per minute
  Day7, Predose: number analyzed (Participants) | 40 | 37
  Day7, Predose | -0.3 [-2.19 to 1.58] | 2.5 [0.55 to 4.39]
  Day7, 0.5 Hour Post-dose: number analyzed (Participants) | 39 | 38
  Day7, 0.5 Hour Post-dose | -0.2 [-2.17 to 1.67] | 3.9 [1.92 to 5.80]
  Day7, 1 Hour Post-dose: number analyzed (Participants) | 39 | 37
  Day7, 1 Hour Post-dose | 0.2 [-1.57 to 1.96] | 4.0 [2.17 to 5.75]
  Day7, 2 Hour Post-dose: number analyzed (Participants) | 40 | 37
  Day7, 2 Hour Post-dose | 1.4 [-0.03 to 2.73] | 2.5 [1.08 to 3.90]
  Day7, 3 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 3 Hour Post-dose | 1.4 [-0.29 to 3.16] | 2.9 [1.15 to 4.65]
  Day7, 3.5 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 3.5 Hour Post-dose | 1.7 [-0.02 to 3.42] | 3.2 [1.41 to 4.90]
  Day7, 4 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 4 Hour Post-dose | 1.1 [-0.68 to 2.86] | 3.3 [1.54 to 5.12]
  Day7, 4.5 Hour Post-dose: number analyzed (Participants) | 40 | 37
  Day7, 4.5 Hour Post-dose | 1.8 [-0.58 to 4.11] | 3.2 [0.80 to 5.58]
  Day7, 5 Hour Post-dose: number analyzed (Participants) | 39 | 36
  Day7, 5 Hour Post-dose | 1.6 [-0.11 to 3.32] | 4.1 [2.33 to 5.82]
  Day7, 6 Hour Post-dose: number analyzed (Participants) | 39 | 37
  Day7, 6 Hour Post-dose | 1.0 [-1.24 to 3.30] | 4.1 [1.81 to 6.41]
  Day7, 8 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 8 Hour Post-dose | 1.1 [-0.90 to 3.05] | 4.2 [2.23 to 6.23]
  Day7, 10 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 10 Hour Post-dose | 0.8 [-1.05 to 2.57] | 5.1 [3.30 to 6.97]
  Day7, 12 Hour Post-dose | 0.4 [-1.56 to 2.44] | 1.1 [-0.92 to 3.11]
  Day7, 24 Hour Post-dose: number analyzed (Participants) | 39 | 36
  Day7, 24 Hour Post-dose | 2.6 [0.70 to 4.53] | 3.9 [1.93 to 5.84]

48. Secondary Outcome: Part 2: Placebo-corrected Change From Baseline in PR Following Administration of GSK3640254 100 mg and GSK3640254 500 mg
Description: Twelve-lead ECGs were recorded in participant using an automated ECG machine. Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Baseline is defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value. Placebo-corrected change from Baseline in PR was calculated as model-predicted mean change from Baseline in PR interval in GSK3640254 group minus model-predicted mean change from Baseline in PR interval in the placebo group.
Time Frame: Baseline (Pre-dose, Day 1) Day 7: Predose and 0.5, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 Hours post dose
Population: QT/QTc Population. Only those participants with data available at the specified time points were analyzed. This outcome measure is intended to provide Placebo-corrected data. Placebo and treatment wise change from Baseline data is provided in outcome measure number 44.
Measure: Least Squares Mean (90% Confidence Interval); unit: Milliseconds
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 40 | 39
Milliseconds
  Day7, Predose: number analyzed (Participants) | 40 | 37
  Day7, Predose | 1.5 [-1.17 to 4.08] | 2.1 [-0.61 to 4.73]
  Day7, 0.5 Hour Post-dose: number analyzed (Participants) | 39 | 38
  Day7, 0.5 Hour Post-dose | 0.4 [-2.33 to 3.10] | 2.5 [-0.27 to 5.22]
  Day7, 1 Hour Post-dose: number analyzed (Participants) | 39 | 37
  Day7, 1 Hour Post-dose | 1.2 [-1.31 to 3.63] | 0.1 [-2.37 to 2.63]
  Day7, 2 Hour Post-dose: number analyzed (Participants) | 40 | 37
  Day7, 2 Hour Post-dose | -0.8 [-2.76 to 1.15] | 1.6 [-0.44 to 3.54]
  Day7, 3 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 3 Hour Post-dose | 0.4 [-1.93 to 2.74] | 2.0 [-0.33 to 4.40]
  Day7, 3.5 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 3.5 Hour Post-dose | 0.9 [-1.44 to 3.20] | 3.2 [0.86 to 5.57]
  Day7, 4 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 4 Hour Post-dose | 1.2 [-0.84 to 3.30] | 1.7 [-0.42 to 3.79]
  Day7, 4.5 Hour Post-dose: number analyzed (Participants) | 40 | 37
  Day7, 4.5 Hour Post-dose | 0.7 [-1.72 to 3.04] | 1.1 [-1.35 to 3.50]
  Day7, 5 Hour Post-dose: number analyzed (Participants) | 39 | 36
  Day7, 5 Hour Post-dose | 0.0 [-2.12 to 2.20] | 0.3 [-1.93 to 2.47]
  Day7, 6 Hour Post-dose: number analyzed (Participants) | 39 | 37
  Day7, 6 Hour Post-dose | 0.2 [-2.22 to 2.70] | 0.2 [-2.30 to 2.69]
  Day7, 8 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 8 Hour Post-dose | -0.3 [-2.57 to 1.91] | 1.1 [-1.13 to 3.41]
  Day7, 10 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 10 Hour Post-dose | 1.1 [-1.00 to 3.13] | 1.1 [-1.00 to 3.18]
  Day7, 12 Hour Post-dose | 0.6 [-1.46 to 2.61] | 1.8 [-0.24 to 3.86]
  Day7, 24 Hour Post-dose: number analyzed (Participants) | 39 | 36
  Day7, 24 Hour Post-dose | -1.4 [-3.58 to 0.69] | -1.8 [-4.00 to 0.36]

49. Secondary Outcome: Part 2: Placebo-corrected Change From Baseline in QRS Following Administration of GSK3640254 100 mg and GSK3640254 500 mg
Description: Twelve-lead ECGs were recorded in participant using an automated ECG machine. Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value. Placebo-corrected change from Baseline in QRS was calculated as model-predicted mean change from Baseline in QRS interval in GSK3640254 group minus model-predicted mean change from Baseline in QRS interval in the placebo group.
Time Frame: Baseline (Pre-dose, Day 1) Day 7: Predose and 0.5, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 Hours post dose
Population: QT/QTc Population. Only those participants with data available at the specified time points were analyzed. This outcome measure is intended to provide Placebo-corrected data. Placebo and treatment wise change from Baseline data is provided in outcome measure number 45.
Measure: Least Squares Mean (90% Confidence Interval); unit: Milliseconds
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 40 | 39
Milliseconds
  Day7, Predose: number analyzed (Participants) | 40 | 37
  Day7, Predose | 0.1 [-0.66 to 0.83] | 0.6 [-0.14 to 1.37]
  Day7, 0.5 Hour Post-dose: number analyzed (Participants) | 39 | 38
  Day7, 0.5 Hour Post-dose | 0.2 [-0.54 to 0.95] | 0.5 [-0.21 to 1.30]
  Day7, 1 Hour Post-dose: number analyzed (Participants) | 39 | 37
  Day7, 1 Hour Post-dose | 0.3 [-0.37 to 1.06] | 0.7 [-0.04 to 1.41]
  Day7, 2 Hour Post-dose: number analyzed (Participants) | 40 | 37
  Day7, 2 Hour Post-dose | 0.5 [-0.26 to 1.20] | 0.7 [-0.04 to 1.44]
  Day7, 3 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 3 Hour Post-dose | 0.5 [-0.18 to 1.24] | 0.4 [-0.29 to 1.15]
  Day7, 3.5 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 3.5 Hour Post-dose | 0.3 [-0.44 to 1.12] | 0.6 [-0.17 to 1.40]
  Day7, 4 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 4 Hour Post-dose | 0.3 [-0.46 to 1.08] | 0.5 [-0.26 to 1.29]
  Day7, 4.5 Hour Post-dose: number analyzed (Participants) | 40 | 37
  Day7, 4.5 Hour Post-dose | 0.2 [-0.59 to 0.97] | 0.4 [-0.40 to 1.18]
  Day7, 5 Hour Post-dose: number analyzed (Participants) | 39 | 36
  Day7, 5 Hour Post-dose | 0.2 [-0.60 to 1.06] | 0.4 [-0.40 to 1.28]
  Day7, 6 Hour Post-dose: number analyzed (Participants) | 39 | 37
  Day7, 6 Hour Post-dose | 0.1 [-0.82 to 1.06] | 0.2 [-0.79 to 1.11]
  Day7, 8 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 8 Hour Post-dose | 0.3 [-0.61 to 1.18] | 0.7 [-0.23 to 1.58]
  Day7, 10 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day7, 10 Hour Post-dose | 0.5 [-0.35 to 1.31] | 0.6 [-0.21 to 1.47]
  Day7, 12 Hour Post-dose | 0.6 [-0.27 to 1.39] | 0.5 [-0.38 to 1.29]
  Day7, 24 Hour Post-dose: number analyzed (Participants) | 39 | 36
  Day7, 24 Hour Post-dose | 0.9 [-0.06 to 1.79] | 1.4 [0.43 to 2.30]

50. Secondary Outcome: Part 2: Number of Participants With Outlier Results for HR, QTcF, ΔQTcF, PR Interval and QRS Interval for GSK3640254 100 mg and GSK3640254 500 mg
Description: Twelve-lead ECGs were recorded using an automated ECG machine with participant in a supine position after a rest of at least 10 minutes. Number of participants with outlier results for HR, QTcF, ΔQTcF, PR interval and QRS interval were summarized.Categorical outlier criteria was as follows:change from Baseline in QTcF (ΔQTcF) >60 ms: Increase of QTc from Baseline > 60 ms, QTcF > 500 ms:Treatment-emergent value of > 500 ms when not present at Baseline (new onset), HR < 50 bpm with a decrease in change from Baseline in heart rate (ΔHR) > 25%:Decrease of HR from Baseline >25% resulting in HR < 50 bpm, HR > 100 bpm with an increase in ΔHR > 25% :Increase of HR from Baseline >25% resulting in HR > 100 bpm, PR > 200 ms with an increase in change from Baseline in PR interval (ΔPR) > 25%:Increase of PR from Baseline > 25% resulting in PR > 200 ms, QRS > 120 ms with an increase in change from Baseline in QRS interval (ΔQRS) > 25%:Increase of QRS from Baseline > 25% resulting in QRS > 120 ms.
Time Frame: Up to Day 51
Population: QT/QTc Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 40 | 39
Participants
  ΔQTcF >60 ms | 0 | 0
  QTcF >500 ms | 0 | 0
  HR <50 bpm with a decrease in ΔHR > 25% | 0 | 0
  HR >100 bpm with an increase in ΔHR > 25% | 1 | 1
  PR >200 ms with an increase in ΔPR > 25% | 0 | 0
  QRS >120 ms an increase in ΔQRS > 25% | 0 | 0

51. Secondary Outcome: Part 2: Number of Participants With Treatment Emergent Changes of T-wave Morphology and Presence of U-wave Following Administration of GSK3640254 100 mg and GSK3640254 500 mg
Description: Twelve-lead ECGs were recorded using an automated ECG machine. Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Flat T-wave=T-amplitude < 1 mm (either positive [+] or negative [-]), including flat isoelectric line, Notched T-wave (+)=Presence of notch(es) of at least 0.05 millivolt (mV) amplitude on ascending or descending arm of the positive T-wave, Biphasic= T-wave that contains a second component with an opposite phase that is at least 0.1 mV deep (both positive/negative and negative/positive and polyphasic T-waves included), Normal T-wave (-)=T-amplitude that is negative, without biphasic T-wave or notches, Notched T-wave (-): Presence of notch(es) of at least 0.05 mV amplitude on descending or ascending arm of the negative T-wave, U-waves= Presence of abnormal U-waves. Data has been reported for Flat T-wave, Notched T-wave (Positive), Biphasic, Normal T-wave (Negative), Notched T-wave (Negative) and T-U wave Fusion.
Time Frame: Up to Day 51
Population: QT/QTc Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 40 | 39
Participants
  Flat T-wave | 2 | 1
  Notched T-wave (Positive) | 0 | 0
  Biphasic | 1 | 0
  Normal T-wave (Negative) | 0 | 0
  Notched T-wave (Negative) | 0 | 0
  T-U wave Fusion | 0 | 0

52. Secondary Outcome: Part 2: Placebo-corrected Change From Baseline in QTcF Following Administration of Moxifloxacin
Description: Twelve-lead ECGs were recorded in participant using an automated ECG machine. Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Baseline is defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value. Placebo-corrected change from Baseline in QTcF was calculated as model-predicted mean change from Baseline in QTcF in moxifloxacin group minus model-predicted mean change from Baseline in QTcF in the placebo group.
Time Frame: Baseline (Pre-dose, Day 1), Day 7: Predose and 0.5, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 Hours post dose
Population: QT/QTc Population. Only those participants with data available at specified time points were analyzed. This outcome measure is intended to provide Placebo-corrected data. Placebo and treatment wise change from Baseline data is provided in outcome measure number 91.
Measure: Least Squares Mean (90% Confidence Interval); unit: Milliseconds
Groups:
- Part 2: Moxifloxacin 400 mg: Participants received placebo matching GSK3640254 from Days 1 through 6 and a single dose of Moxifloxacin 400 mg on Day 7 in each Treatment Period of Part 2 of the study.
Arm/Group | Part 2: Moxifloxacin 400 mg
Number analyzed (Participants) | 40
Milliseconds
  Day 7, Predose | 0.6 [-1.74 to 2.90]
  Day7, 0.5 Hour Post-dose | -0.2 [-2.82 to 2.37]
  Day 7, 1 Hour Post-dose | -0.8 [-3.50 to 1.88]
  Day7, 2 Hour Post-dose | 5.6 [2.57 to 8.61]
  Day 7, 3 Hour Post-dose | 7.9 [4.94 to 10.92]
  Day7, 3.5 Hour Post-dose | 8.9 [6.15 to 11.60]
  Day7, 4 Hour Post-dose | 8.6 [6.07 to 11.21]
  Day7, 4.5 Hour Post-dose | 8.4 [5.62 to 11.18]
  Day7, 5 Hour Post-dose | 8.2 [5.53 to 10.79]
  Day7, 6 Hour Post-dose | 8.2 [4.94 to 11.50]
  Day7, 8 Hour Post-dose | 6.9 [4.19 to 9.66]
  Day7, 10 Hour Post-dose | 6.8 [4.30 to 9.28]
  Day7, 12 Hour Post-dose | 5.3 [2.38 to 8.17]
  Day7, 24 Hour Post-dose | 6.8 [4.13 to 9.54]

53. Secondary Outcome: Part 2: AUC(0-t) of GSK3640254 100 mg and GSK3640254 500 mg
Description: Blood samples were collected at indicated time points. PK analysis was conducted using standard non-compartmental methods .
Time Frame: as for outcome 40
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 40 | 40
Hours*nanograms per milliliter | 13840 (37.2) | 67520 (42.9)

54. Secondary Outcome: Part 2: AUC(0-tau) of GSK3640254 100 mg and GSK3640254 500 mg
Description: as for outcome 2
Time Frame: as for outcome 40
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 40 | 40
Hours*nanograms per milliliter | 13830 (37.2) | 67490 (42.9)

55. Secondary Outcome: Part 2: Cmax of GSK3640254 100 mg and GSK3640254 500 mg
Description: as for outcome 2
Time Frame: as for outcome 40
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 40 | 40
Nanograms per milliliter | 830.3 (37.9) | 4261 (41.8)

56. Secondary Outcome: Part 2: Ctau of GSK3640254 100 mg and GSK3640254 500 mg
Description: as for outcome 2
Time Frame: as for outcome 40
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 40 | 40
Nanograms per milliliter | 459.9 (40.3) | 2137 (46.6)

57. Secondary Outcome: Part 2: Tmax of GSK3640254 100 mg and GSK3640254 500 mg
Description: as for outcome 2
Time Frame: as for outcome 40
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 40 | 40
Hours | 5.008 [2.07 to 12.00] | 5.000 [2.00 to 12.00]

58. Secondary Outcome: Part 2: Cmax of Moxifloxacin 400 mg
Description: as for outcome 2
Time Frame: as for outcome 40
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 2: Moxifloxacin 400 mg
Number analyzed (Participants) | 40
Nanograms per milliliter | 1964 (20.2)

59. Secondary Outcome: Part 2: Tmax of Moxifloxacin 400 mg
Description: as for outcome 2
Time Frame: as for outcome 40
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Moxifloxacin 400 mg
Number analyzed (Participants) | 40
Hours | 4.000 [2.00 to 6.00]

60. Secondary Outcome: Part 2: Number of Participants With Non-SAEs and SAEs
Description: as for outcome 8
Time Frame: Up to Day 51
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Participants
  Non SAE | 7 | 4 | 5 | 10
  SAE | 0 | 0 | 0 | 0

61. Secondary Outcome: Part 2: Absolute Values for Hematology Parameter: Hemoglobin
Description: Blood samples were collected at indicated time points to analyze hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Grams per liter
  Baseline (Day -2) | 141.8 (12.90) | 140.5 (15.05) | 141.6 (15.47) | 141.7 (14.37)
  Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Day 8 | 139.9 (14.26) | 140.3 (13.45) | 140.4 (14.81) | 143.4 (15.00)
  Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Day 9 | 139.4 (18.82) | 140.0 (13.60) | 143.7 (10.15) | 137.7 (11.49)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Day 14 | 140.7 (14.01) | 140.1 (12.91) | 142.1 (16.28) | 142.2 (15.27)

62. Secondary Outcome: Part 2: Absolute Values for Hematology Parameter: Hematocrit
Description: Blood samples were collected at indicated time points to analyze hematocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits
Time Frame: Baseline (Day -2), Day 8, Day 9, Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Proportion of red blood cells in blood
  Baseline (Day -2) | 0.4163 (0.03226) | 0.4131 (0.03985) | 0.4157 (0.04031) | 0.4167 (0.03829)
  Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Day 8 | 0.4099 (0.03700) | 0.4120 (0.03334) | 0.4123 (0.03874) | 0.4171 (0.03831)
  Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Day 9 | 0.4134 (0.04315) | 0.4086 (0.03431) | 0.4247 (0.02835) | 0.4029 (0.03272)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Day 14 | 0.4118 (0.03753) | 0.4107 (0.03242) | 0.4175 (0.04266) | 0.4189 (0.03960)

63. Secondary Outcome: Part 2: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected at indicated time points to analyze erythrocytes mean corpuscular volume. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits
Time Frame: Baseline (Day -2), Day 8, Day 9, Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Femtoliter
  Baseline (Day -2) | 85.93 (5.041) | 85.96 (5.039) | 86.26 (4.971) | 85.92 (4.767)
  Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Day 8 | 85.95 (3.851) | 85.57 (5.391) | 86.29 (5.417) | 84.91 (4.948)
  Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Day 9 | 85.00 (7.113) | 86.42 (3.592) | 84.61 (2.623) | 87.08 (4.109)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Day 14 | 86.25 (3.841) | 86.17 (5.378) | 86.05 (5.265) | 85.53 (4.993)

64. Secondary Outcome: Part 2: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected at indicated time points to analyze erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 8, Day 9, Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Picograms
  Baseline (Day -2) | 29.27 (2.308) | 29.23 (2.077) | 29.37 (2.062) | 29.21 (2.005)
  Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Day 8 | 29.34 (1.603) | 29.13 (2.325) | 29.39 (2.273) | 29.17 (2.189)
  Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Day 9 | 28.67 (3.417) | 29.56 (1.551) | 28.62 (1.362) | 29.79 (1.516)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Day 14 | 29.45 (1.487) | 29.40 (2.449) | 29.29 (2.227) | 29.02 (2.137)

65. Secondary Outcome: Part 2: Absolute Values for Hematology Parameter: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets and Leukocytes
Description: Blood samples were collected at indicated time points to analyze basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelets and leukocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 8, Day 9, Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
10^9 cells per liter
  Basophils,Baseline (Day -2) | 0.035 (0.0194) | 0.036 (0.0228) | 0.037 (0.0218) | 0.031 (0.0121)
  Basophils,Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Basophils,Day 8 | 0.035 (0.0228) | 0.032 (0.0176) | 0.030 (0.0149) | 0.039 (0.0157)
  Basophils,Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Basophils,Day 9 | 0.032 (0.0155) | 0.036 (0.0191) | 0.039 (0.0145) | 0.025 (0.0108)
  Basophils,Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Basophils,Day 14 | 0.033 (0.0178) | 0.031 (0.0161) | 0.033 (0.0177) | 0.040 (0.0242)
  Eosinophils,Baseline (Day -2) | 0.124 (0.0775) | 0.127 (0.0794) | 0.135 (0.0966) | 0.123 (0.0716)
  Eosinophils,Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Eosinophils,Day 8 | 0.116 (0.0637) | 0.136 (0.0757) | 0.130 (0.0797) | 0.135 (0.0725)
  Eosinophils,Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Eosinophils,Day 9 | 0.167 (0.0859) | 0.120 (0.0754) | 0.114 (0.0688) | 0.081 (0.0418)
  Eosinophils,Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Eosinophils,Day 14 | 0.113 (0.0765) | 0.131 (0.0918) | 0.126 (0.0717) | 0.141 (0.0737)
  Lymphocytes,Baseline (Day -2) | 1.694 (0.5355) | 1.830 (0.5683) | 1.736 (0.5498) | 1.677 (0.4789)
  Lymphocytes,Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Lymphocytes,Day 8 | 1.641 (0.4661) | 1.605 (0.4496) | 1.675 (0.5013) | 1.688 (0.4620)
  Lymphocytes,Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Lymphocytes,Day 9 | 1.603 (0.2137) | 1.907 (0.6142) | 1.637 (0.5265) | 1.540 (0.5550)
  Lymphocytes,Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Lymphocytes,Day 14 | 1.710 (0.5906) | 1.606 (0.5602) | 1.705 (0.4747) | 1.755 (0.5892)
  Monocytes,Baseline (Day -2) | 0.427 (0.1533) | 0.442 (0.1429) | 0.451 (0.1588) | 0.429 (0.1476)
  Monocytes,Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Monocytes,Day 8 | 0.426 (0.1090) | 0.436 (0.1518) | 0.456 (0.1521) | 0.501 (0.1609)
  Monocytes,Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Monocytes,Day 9 | 0.485 (0.1499) | 0.468 (0.1376) | 0.389 (0.1312) | 0.350 (0.1040)
  Monocytes,Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Monocytes,Day 14 | 0.413 (0.1474) | 0.399 (0.1469) | 0.431 (0.1514) | 0.448 (0.1402)
  Neutrophils, Baseline (Day -2) | 2.842 (0.9011) | 2.902 (0.8438) | 2.957 (1.0517) | 2.829 (0.8172)
  Neutrophils,Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Neutrophils,Day 8 | 2.889 (0.9751) | 2.671 (0.8247) | 2.825 (0.8364) | 2.952 (0.9562)
  Neutrophils,Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Neutrophils,Day 9 | 2.990 (0.9534) | 2.618 (0.8351) | 2.619 (1.1073) | 2.530 (0.5010)
  Neutrophils,Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Neutrophils,Day 14 | 2.712 (0.8786) | 2.506 (0.7270) | 2.758 (0.8062) | 2.750 (0.7833)
  Platelets,Baseline (Day -2) | 233.7 (42.39) | 237.1 (46.09) | 234.0 (48.15) | 230.8 (48.34)
  Platelets, Day 8: number analyzed (Participants) | 31 | 29 | 30 | 28
  Platelets, Day 8 | 228.9 (43.10) | 226.4 (43.06) | 234.8 (47.94) | 224.7 (41.97)
  Platelets, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Platelets, Day 9 | 221.4 (34.16) | 233.3 (62.32) | 225.9 (52.60) | 235.4 (30.80)
  Platelets, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Platelets, Day 14 | 231.6 (48.26) | 227.1 (44.07) | 234.0 (40.87) | 226.7 (46.75)
  Leukocytes, Baseline (Day -2) | 5.12 (1.205) | 5.34 (1.153) | 5.31 (1.325) | 5.08 (1.092)
  Leukocytes,Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Leukocytes,Day 8 | 5.10 (1.223) | 4.87 (0.985) | 5.11 (1.151) | 5.32 (1.172)
  Leukocytes,Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Leukocytes,Day 9 | 5.27 (1.125) | 5.14 (1.307) | 4.78 (1.411) | 4.53 (0.850)
  Leukocytes,Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Leukocytes,Day 14 | 4.97 (1.184) | 4.67 (1.040) | 5.05 (1.054) | 5.14 (1.023)

66. Secondary Outcome: Part 2: Absolute Values for Hematology Parameter: Erythrocytes
Description: Blood samples were collected at indicated time points to analyze Erythrocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
10^12 cells per liter
  Baseline (Day -2) | 4.859 (0.4614) | 4.815 (0.4808) | 4.829 (0.4842) | 4.864 (0.5017)
  Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Day 8 | 4.775 (0.4512) | 4.833 (0.4585) | 4.794 (0.5278) | 4.927 (0.5074)
  Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Day 9 | 4.890 (0.6010) | 4.737 (0.4416) | 5.023 (0.3646) | 4.632 (0.3654)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Day 14 | 4.782 (0.4689) | 4.780 (0.4388) | 4.866 (0.5418) | 4.910 (0.5078)

67. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected at indicated time points to analyze hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Grams per liter
  Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Day 8 | -2.7 (5.58) | 0.1 (6.08) | -0.9 (6.20) | 0.3 (4.45)
  Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Day 9 | -0.6 (5.17) | -1.3 (5.87) | 1.0 (6.54) | 0.0 (4.78)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Day 14 | -1.9 (6.15) | -0.2 (5.43) | 0.8 (7.32) | -0.9 (4.53)

68. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected at indicated time points to analyze hematocrit . Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Proportion of red blood cells in blood
  Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Day 8 | -0.0068 (0.01715) | 0.0002 (0.01915) | -0.0018 (0.01861) | -0.0040 (0.01256)
  Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Day 9 | -0.0009 (0.01290) | -0.0076 (0.01928) | 0.0036 (0.02174) | -0.0007 (0.01843)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Day 14 | -0.0052 (0.01837) | -0.0012 (0.01728) | 0.0035 (0.02158) | -0.0026 (0.01427)

69. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected at indicated time points to analyze erythrocytes mean corpuscular volume. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Femtoliter
  Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Day 8 | -0.57 (2.043) | -0.26 (0.748) | -0.45 (0.720) | -0.55 (2.011)
  Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Day 9 | 0.15 (0.438) | 0.10 (0.559) | -0.01 (0.695) | -0.20 (0.785)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Day 14 | -0.33 (2.255) | 0.35 (2.379) | -0.69 (2.122) | -0.02 (2.074)

70. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected at indicated time points to analyze erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Picograms
  Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Day 8 | -0.25 (1.052) | -0.08 (0.379) | -0.18 (0.417) | 0.15 (1.042)
  Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Day 9 | -0.05 (0.635) | 0.27 (0.469) | -0.06 (0.617) | 0.01 (0.486)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Day 14 | -0.15 (1.188) | 0.19 (1.186) | -0.28 (1.073) | -0.01 (1.113)

71. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets and Leukocytes
Description: Blood samples were collected at indicated time points to analyze basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelets and leukocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
10^9 cells per liter
  Basophils,Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Basophils,Day 8 | -0.002 (0.0141) | -0.003 (0.0111) | -0.004 (0.0088) | 0.005 (0.0107)
  Basophils,Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Basophils,Day 9 | 0.002 (0.0123) | -0.003 (0.0101) | -0.010 (0.0240) | 0.002 (0.0103)
  Basophils,Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Basophils,Day 14 | -0.005 (0.0178) | -0.004 (0.0105) | -0.001 (0.0116) | 0.007 (0.0245)
  Eosinophils,Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Eosinophils,Day 8 | 0.002 (0.0363) | 0.007 (0.0405) | -0.008 (0.0525) | -0.001 (0.0367)
  Eosinophils,Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Eosinophils,Day 9 | 0.008 (0.0339) | -0.004 (0.0347) | -0.011 (0.0285) | -0.002 (0.0204)
  Eosinophils,Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Eosinophils,Day 14 | -0.004 (0.0382) | 0.002 (0.0641) | -0.012 (0.0528) | 0.006 (0.0507)
  Lymphocytes,Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Lymphocytes,Day 8 | -0.129 (0.3091) | -0.161 (0.3238) | -0.071 (0.3535) | -0.039 (0.2684)
  Lymphocytes,Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Lymphocytes,Day 9 | 0.122 (0.1852) | -0.092 (0.3865) | -0.067 (0.2649) | 0.015 (0.2089)
  Lymphocytes,Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Lymphocytes,Day 14 | -0.066 (0.2859) | -0.160 (0.2649) | -0.041 (0.3457) | 0.014 (0.3589)
  Monocytes,Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Monocytes,Day 8 | 0.001 (0.1206) | 0.014 (0.0900) | -0.015 (0.1119) | 0.034 (0.1148)
  Monocytes,Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Monocytes,Day 9 | 0.047 (0.0638) | -0.030 (0.1627) | 0.010 (0.0332) | 0.038 (0.0382)
  Monocytes,Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Monocytes,Day 14 | -0.015 (0.1347) | -0.022 (0.1413) | -0.040 (0.0967) | -0.022 (0.1388)
  Neutrophils,Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Neutrophils,Day 8 | 0.018 (0.8722) | -0.272 (0.6668) | -0.319 (0.7755) | -0.022 (0.7040)
  Neutrophils,Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Neutrophils,Day 9 | 0.332 (0.3485) | -0.174 (0.8246) | 0.306 (0.4508) | 0.136 (0.4495)
  Neutrophils,Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Neutrophils,Day 14 | -0.155 (0.5886) | -0.437 (0.7038) | -0.386 (0.6994) | -0.262 (0.5618)
  Platelets, Day 8: number analyzed (Participants) | 31 | 29 | 30 | 28
  Platelets, Day 8 | -7.4 (23.57) | -10.8 (30.25) | -2.2 (28.56) | -4.5 (24.10)
  Platelets, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Platelets, Day 9 | -8.4 (21.44) | -3.5 (22.10) | 0.7 (25.99) | 7.9 (28.29)
  Platelets, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Platelets, Day 14 | -3.2 (34.31) | -10.1 (31.76) | -2.5 (31.02) | -6.7 (28.80)
  Leukocytes,Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Leukocytes,Day 8 | -0.11 (1.122) | -0.42 (0.858) | -0.41 (0.943) | -0.01 (0.837)
  Leukocytes,Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Leukocytes,Day 9 | 0.50 (0.406) | -0.32 (1.138) | 0.20 (0.505) | 0.21 (0.626)
  Leukocytes,Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Leukocytes,Day 14 | -0.24 (0.669) | -0.63 (0.864) | -0.47 (0.856) | -0.24 (0.721)

72. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected at indicated time points to analyze erythrocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
10^12 cells per liter
  Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Day 8 | -0.049 (0.2246) | 0.022 (0.2160) | 0.008 (0.2079) | -0.015 (0.1855)
  Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Day 9 | -0.023 (0.1546) | -0.090 (0.2291) | 0.044 (0.2637) | 0.004 (0.2052)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Day 14 | -0.043 (0.2695) | -0.031 (0.2130) | 0.081 (0.2488) | -0.031 (0.1956)

73. Secondary Outcome: Part 2: Absolute Values for Chemistry Parameters: Glucose, Cholesterol, Magnesium, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium, Blood Urea Nitrogen
Description: Blood samples were collected at indicated time points to analyze glucose, cholesterol, magnesium, triglycerides, anion gap, calcium, carbon dioxide, chloride, phosphate, potassium, sodium, and blood urea nitrogen. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visit.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Millimoles per liter
  Glucose,Baseline (Day -2) | 4.813 (0.3180) | 4.739 (0.3538) | 4.810 (0.3038) | 4.753 (0.2744)
  Glucose, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Glucose, Day 8 | 4.777 (0.2914) | 4.749 (0.2843) | 4.798 (0.2707) | 4.670 (0.2420)
  Glucose, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Glucose, Day 9 | 4.763 (0.2295) | 4.668 (0.4071) | 4.811 (0.3717) | 4.791 (0.2795)
  Glucose, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Glucose, Day 14 | 4.794 (0.2526) | 4.777 (0.2745) | 4.713 (0.3106) | 4.749 (0.2474)
  Cholesterol, Baseline (Day -2) | 4.323 (0.8707) | 4.330 (0.7859) | 4.243 (0.8603) | 4.350 (0.7624)
  Cholesterol, Day 8,: number analyzed (Participants) | 31 | 29 | 31 | 30
  Cholesterol, Day 8, | 4.300 (0.8340) | 4.246 (0.8197) | 4.147 (0.7439) | 4.186 (0.7233)
  Cholesterol, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Cholesterol, Day 9 | 3.988 (0.5501) | 4.253 (0.8441) | 4.467 (0.8551) | 4.050 (0.7872)
  Cholesterol, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Cholesterol, Day 14 | 4.361 (0.8290) | 4.180 (0.8088) | 4.233 (0.7982) | 4.145 (0.7483)
  Magnesium, Baseline (Day -2) | 0.794 (0.0653) | 0.796 (0.0688) | 0.791 (0.0679) | 0.793 (0.0709)
  Magnesium, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Magnesium, Day 8 | 0.793 (0.0499) | 0.769 (0.0565) | 0.783 (0.0610) | 0.793 (0.0539)
  Magnesium, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Magnesium, Day 9 | 0.736 (0.0610) | 0.820 (0.0400) | 0.771 (0.0521) | 0.817 (0.0736)
  Magnesium, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Magnesium, Day 14 | 0.796 (0.0627) | 0.789 (0.0662) | 0.801 (0.0675) | 0.796 (0.0579)
  Triglycerides, Baseline (Day -2) | 1.011 (0.4865) | 1.059 (0.4907) | 0.996 (0.4214) | 0.978 (0.4082)
  Triglycerides, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Triglycerides, Day 8 | 0.977 (0.4124) | 0.958 (0.4513) | 0.980 (0.3876) | 0.894 (0.3583)
  Triglycerides, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Triglycerides, Day 9 | 1.036 (0.4571) | 0.935 (0.2874) | 0.891 (0.3760) | 0.778 (0.4061)
  Triglycerides, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Triglycerides, Day 14 | 0.948 (0.3862) | 0.941 (0.3983) | 1.013 (0.4432) | 1.049 (0.3844)
  Anion gap, Baseline (Day -2) | 10.0 (1.46) | 10.2 (1.42) | 9.9 (1.61) | 10.5 (1.65)
  Anion gap, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Anion gap, Day 8 | 10.1 (1.41) | 10.3 (1.20) | 10.1 (1.44) | 10.1 (1.41)
  Anion gap, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Anion gap, Day 9 | 10.0 (1.56) | 11.1 (1.64) | 10.8 (1.30) | 10.8 (1.69)
  Anion gap, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Anion gap, Day 14 | 9.9 (1.36) | 9.9 (1.36) | 10.2 (1.42) | 9.8 (1.35)
  Calcium, Baseline (Day -2) | 2.371 (0.0868) | 2.363 (0.0942) | 2.350 (0.0939) | 2.375 (0.0922)
  Calcium, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Calcium, Day 8 | 2.317 (0.0920) | 2.316 (0.0893) | 2.316 (0.0876) | 2.316 (0.0945)
  Calcium, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Calcium, Day 9 | 2.357 (0.0793) | 2.366 (0.0595) | 2.402 (0.0978) | 2.332 (0.0627)
  Calcium, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Calcium, Day 14 | 2.367 (0.0913) | 2.349 (0.0802) | 2.391 (0.0918) | 2.358 (0.1040)
  Carbon dioxide, Baseline (Day -2) | 30.4 (2.08) | 30.2 (1.42) | 30.5 (1.58) | 30.2 (2.07)
  Carbon dioxide, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Carbon dioxide, Day 8 | 29.3 (2.32) | 29.6 (1.76) | 29.2 (1.63) | 29.3 (1.95)
  Carbon dioxide, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Carbon dioxide, Day 9 | 30.2 (1.55) | 29.2 (1.54) | 30.0 (2.18) | 28.9 (2.13)
  Carbon dioxide, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Carbon dioxide, Day 14 | 30.3 (1.84) | 30.3 (1.85) | 30.5 (1.82) | 30.8 (1.68)
  Chloride, Baseline (Day -2) | 102.8 (1.57) | 103.4 (1.87) | 103.3 (2.05) | 103.2 (1.98)
  Chloride, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Chloride, Day 8 | 103.5 (1.91) | 102.6 (1.61) | 103.0 (1.64) | 102.5 (1.80)
  Chloride, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Chloride, Day 9 | 102.4 (1.51) | 103.9 (1.76) | 102.8 (1.72) | 103.0 (1.63)
  Chloride, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Chloride, Day 14 | 103.9 (1.77) | 103.3 (1.34) | 103.6 (1.70) | 103.5 (1.74)
  Phosphate, Baseline (Day -2) | 1.190 (0.1394) | 1.199 (0.1552) | 1.182 (0.1550) | 1.172 (0.1686)
  Phosphate, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Phosphate, Day 8 | 1.194 (0.1272) | 1.195 (0.1410) | 1.186 (0.1408) | 1.168 (0.1644)
  Phosphate, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Phosphate, Day 9 | 1.166 (0.1436) | 1.292 (0.1254) | 1.212 (0.1213) | 1.193 (0.1076)
  Phosphate, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Phosphate, Day 14 | 1.233 (0.1450) | 1.164 (0.1264) | 1.222 (0.1415) | 1.219 (0.1625)
  Potassium, Baseline (Day -2) | 4.30 (0.337) | 4.34 (0.327) | 4.35 (0.315) | 4.32 (0.331)
  Potassium, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Potassium, Day 8 | 4.29 (0.291) | 4.26 (0.324) | 4.20 (0.275) | 4.07 (0.296)
  Potassium, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Potassium, Day 9 | 4.26 (0.222) | 4.17 (0.310) | 4.42 (0.484) | 4.18 (0.416)
  Potassium, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Potassium, Day 14 | 4.39 (0.389) | 4.41 (0.232) | 4.43 (0.301) | 4.44 (0.337)
  Sodium, Baseline (Day -2) | 138.8 (1.91) | 139.4 (1.80) | 139.2 (2.18) | 139.4 (1.51)
  Sodium, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Sodium, Day 8 | 138.6 (1.89) | 138.2 (1.55) | 138.1 (1.25) | 137.8 (1.70)
  Sodium, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Sodium, Day 9 | 138.4 (0.70) | 139.9 (2.21) | 139.2 (1.39) | 138.6 (1.43)
  Sodium, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Sodium, Day 14 | 139.6 (1.65) | 139.0 (1.61) | 139.9 (1.20) | 139.6 (2.01)
  Blood Urea Nitrogen, Baseline(Day-2) | 4.325 (1.0398) | 4.419 (0.9822) | 4.573 (1.3349) | 4.414 (1.2366)
  Blood Urea Nitrogen, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Blood Urea Nitrogen, Day 8 | 5.242 (0.9369) | 5.156 (1.0329) | 4.805 (0.8952) | 4.675 (0.9487)
  Blood Urea Nitrogen, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Blood Urea Nitrogen, Day 9 | 4.472 (0.5020) | 5.453 (0.9684) | 5.251 (0.6649) | 4.243 (0.8860)
  Blood Urea Nitrogen, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Blood Urea Nitrogen, Day 14 | 4.637 (0.7997) | 4.440 (0.9129) | 4.428 (0.9272) | 4.451 (0.9627)

74. Secondary Outcome: Part 2: Absolute Values for Chemistry Parameters: ALT, ALP, AST, GGT, Creatine Kinase, Lactate Dehydrogenase
Description: Blood samples were collected at indicated time points to analyze ALT, ALP, AST, GGT, creatine kinase, and lactate dehydrogenase. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visit.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
International units per liter
  ALT, Baseline (Day -2) | 18.3 (10.92) | 16.8 (10.26) | 17.5 (10.40) | 16.3 (9.35)
  ALT, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  ALT, Day 8 | 14.0 (7.46) | 17.2 (9.80) | 15.7 (10.63) | 19.5 (11.46)
  ALT, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  ALT, Day 9 | 26.6 (16.04) | 12.5 (9.50) | 14.2 (4.29) | 16.4 (8.69)
  ALT, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  ALT, Day 14 | 13.8 (6.38) | 18.7 (12.07) | 16.6 (11.05) | 19.0 (11.34)
  ALP, Baseline (Day -2) | 58.7 (13.67) | 58.3 (13.52) | 58.0 (13.82) | 58.9 (14.23)
  ALP, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  ALP, Day 8 | 56.8 (11.95) | 55.6 (12.06) | 57.1 (12.81) | 59.6 (13.52)
  ALP, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  ALP, Day 9 | 56.1 (15.32) | 63.5 (15.28) | 58.9 (12.64) | 53.0 (8.03)
  ALP, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  ALP, Day 14 | 56.7 (13.21) | 55.1 (10.80) | 58.8 (13.98) | 59.4 (14.15)
  AST, Baseline (Day -2) | 15.8 (4.73) | 15.5 (4.56) | 15.5 (3.78) | 15.3 (3.88)
  AST, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  AST, Day 8 | 14.0 (3.18) | 16.0 (9.92) | 13.7 (3.14) | 15.6 (4.01)
  AST, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  AST, Day 9 | 17.3 (5.14) | 13.6 (3.26) | 15.6 (5.05) | 15.1 (3.75)
  AST, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  AST, Day 14 | 14.1 (3.10) | 15.3 (3.81) | 14.5 (3.96) | 15.8 (5.22)
  GGT, Baseline (Day -2) | 16.7 (11.06) | 17.2 (11.41) | 16.6 (8.75) | 16.7 (10.53)
  GGT, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  GGT, Day 8 | 15.0 (11.16) | 17.9 (11.53) | 15.2 (7.30) | 18.7 (10.22)
  GGT, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  GGT, Day 9 | 20.3 (7.63) | 12.5 (6.56) | 19.1 (11.61) | 10.8 (2.44)
  GGT, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  GGT, Day 14 | 14.7 (10.48) | 17.5 (12.44) | 15.1 (7.28) | 17.7 (9.01)
  Creatine kinase, Baseline (Day -2) | 103.0 (61.10) | 120.8 (95.60) | 112.6 (91.50) | 117.8 (105.69)
  Creatine kinase, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Creatine kinase, Day 8 | 72.8 (42.00) | 163.9 (428.51) | 82.5 (48.77) | 90.3 (51.09)
  Creatine kinase, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Creatine kinase, Day 9 | 173.4 (136.99) | 75.5 (45.25) | 171.1 (184.31) | 81.1 (40.14)
  Creatine kinase, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Creatine kinase, Day 14 | 102.1 (113.21) | 104.9 (63.56) | 91.7 (55.00) | 110.1 (76.61)
  Lactatedehydrogenase, Baseline(Day-2) | 119.9 (21.33) | 122.8 (21.04) | 119.6 (18.16) | 121.2 (24.03)
  Lactate dehydrogenase, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Lactate dehydrogenase, Day 8 | 107.5 (18.24) | 111.8 (19.37) | 108.0 (17.13) | 113.5 (16.87)
  Lactate dehydrogenase, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Lactate dehydrogenase, Day 9 | 124.0 (20.88) | 107.4 (20.66) | 118.2 (16.69) | 108.1 (17.01)
  Lactate dehydrogenase, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Lactate dehydrogenase, Day 14 | 113.4 (17.68) | 113.5 (17.09) | 116.6 (18.19) | 118.8 (20.87)

75. Secondary Outcome: Part 2: Absolute Values for Chemistry Parameters: Creatinine, Urate, Total Bilirubin, Direct Bilirubin
Description: Blood samples were collected at indicated timepoints to analyze creatinine, urate, total bilirubin, and direct bilirubin. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visit.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Micromoles per liter
  Creatinine, Baseline (Day -2) | 80.51 (13.855) | 79.38 (14.340) | 81.86 (14.819) | 79.83 (14.976)
  Creatinine, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Creatinine, Day 8 | 78.45 (16.058) | 88.55 (16.380) | 78.38 (15.118) | 82.01 (16.558)
  Creatinine, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Creatinine, Day 9 | 86.89 (13.446) | 77.07 (17.015) | 89.38 (14.323) | 80.63 (15.048)
  Creatinine, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Creatinine, Day 14 | 79.56 (16.792) | 84.19 (13.996) | 79.16 (15.043) | 81.47 (14.487)
  Urate, Baseline (Day -2) | 297.5 (60.11) | 294.6 (57.22) | 293.6 (62.59) | 295.3 (59.89)
  Urate, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Urate, Day 8 | 288.3 (53.21) | 302.1 (51.50) | 286.7 (58.76) | 277.6 (58.06)
  Urate, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Urate, Day 9 | 290.2 (64.04) | 295.3 (55.91) | 307.2 (46.23) | 261.1 (50.55)
  Urate, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Urate, Day 14 | 291.4 (49.07) | 293.1 (54.91) | 290.1 (56.69) | 285.4 (56.39)
  Total Bilirubin, Baseline (Day -2) | 12.18 (6.249) | 11.79 (5.406) | 11.13 (4.812) | 11.79 (4.654)
  Total Bilirubin, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Total Bilirubin, Day 8 | 9.91 (3.647) | 10.36 (4.712) | 10.68 (4.792) | 11.63 (4.090)
  Total Bilirubin, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Total Bilirubin, Day 9 | 12.50 (6.712) | 13.71 (2.889) | 13.16 (6.586) | 12.00 (4.901)
  Total Bilirubin, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Total Bilirubin, Day 14 | 11.42 (4.666) | 12.89 (7.360) | 12.40 (5.214) | 11.53 (4.675)
  Direct Bilirubin, Baseline (Day -2) | 2.22 (0.988) | 2.12 (0.916) | 2.05 (0.834) | 2.07 (0.686)
  Direct Bilirubin, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Direct Bilirubin, Day 8 | 1.86 (0.689) | 1.90 (0.796) | 1.97 (0.811) | 2.22 (0.934)
  Direct Bilirubin, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Direct Bilirubin, Day 9 | 2.23 (1.033) | 2.39 (0.646) | 2.30 (1.127) | 2.23 (0.772)
  Direct Bilirubin, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Direct Bilirubin, Day 14 | 2.06 (0.781) | 2.21 (1.113) | 2.22 (0.887) | 2.10 (0.844)

76. Secondary Outcome: Part 2: Absolute Values for Chemistry Parameters: Albumin, Globulin, Total Protein
Description: Blood samples were collected at indicated timepoints to analyze albumin, globulin, and total protein. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visit.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Grams per liter
  Albumin, Baseline (Day -2) | 43.8 (2.89) | 44.0 (3.12) | 43.6 (3.18) | 44.5 (3.33)
  Albumin, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Albumin, Day 8 | 41.7 (2.86) | 42.0 (3.39) | 42.2 (2.55) | 42.8 (2.57)
  Albumin, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Albumin, Day 9 | 42.7 (2.83) | 43.5 (1.63) | 44.0 (3.28) | 43.5 (2.59)
  Albumin, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Albumin, Day 14 | 43.2 (2.96) | 42.8 (2.68) | 43.9 (3.20) | 42.8 (2.59)
  Globulin, Baseline (Day -2) | 26.6 (4.43) | 26.0 (3.77) | 25.9 (3.99) | 26.3 (3.58)
  Globulin, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Globulin, Day 8 | 25.1 (4.04) | 26.4 (3.89) | 25.5 (4.06) | 26.4 (3.51)
  Globulin, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Globulin, Day 9 | 29.3 (1.89) | 24.5 (3.01) | 26.9 (3.89) | 25.6 (3.86)
  Globulin, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Globulin, Day 14 | 25.0 (3.33) | 26.6 (3.88) | 26.4 (4.21) | 26.1 (3.84)
  Total protein, Baseline (Day -2) | 70.4 (5.22) | 70.0 (4.69) | 69.5 (4.55) | 70.7 (5.02)
  Total protein, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Total protein, Day 8 | 66.8 (4.09) | 68.4 (4.70) | 67.8 (4.31) | 69.2 (4.11)
  Total protein, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Total protein, Day 9 | 72.0 (3.09) | 67.9 (3.83) | 70.9 (4.14) | 69.1 (4.15)
  Total protein, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Total protein, Day 14 | 68.2 (4.26) | 69.4 (3.80) | 70.3 (5.01) | 68.8 (5.09)

77. Secondary Outcome: Part 2: Absolute Values for Chemistry Parameters: Amylase and Lipase
Description: Blood samples were collected at indicated timepoints to analyze amylase and lipase. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visit.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Units per liter
  Amylase, Baseline (Day -2) | 55.7 (21.74) | 55.9 (22.19) | 58.2 (24.65) | 56.2 (25.45)
  Amylase, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Amylase, Day 8 | 52.4 (21.70) | 59.1 (26.80) | 53.4 (19.71) | 57.7 (22.34)
  Amylase, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Amylase, Day 9 | 66.3 (19.41) | 49.2 (16.70) | 61.0 (26.37) | 44.6 (17.40)
  Amylase, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Amylase, Day 14 | 50.9 (20.92) | 58.5 (24.58) | 52.9 (20.11) | 58.0 (21.02)
  Lipase, Baseline (Day -2), | 25.3 (10.98) | 26.5 (11.59) | 27.0 (11.06) | 27.5 (13.93)
  Lipase, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Lipase, Day 8 | 29.3 (27.50) | 26.5 (12.22) | 25.2 (12.39) | 26.6 (12.87)
  Lipase, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Lipase, Day 9 | 28.4 (12.99) | 23.7 (10.47) | 28.1 (12.26) | 22.7 (6.99)
  Lipase, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Lipase, Day 14 | 23.6 (9.21) | 26.7 (10.84) | 24.8 (9.45) | 26.6 (11.79)

78. Secondary Outcome: Part 2: Change From Baseline in Chemistry Parameters: Glucose, Cholesterol, Magnesium, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium, Blood Urea Nitrogen
Description: Blood samples were collected at indicated time points to analyze glucose, cholesterol, magnesium, triglycerides, anion gap, calcium, carbon dioxide, chloride, phosphate, potassium, sodium, and blood urea nitrogen.Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visit. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Millimoles per liter
  Glucose, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Glucose, Day 8 | -0.041 (0.2820) | 0.029 (0.3396) | -0.023 (0.3001) | -0.024 (0.2263)
  Glucose, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Glucose, Day 9 | 0.023 (0.3045) | -0.119 (0.3171) | 0.040 (0.1949) | -0.139 (0.2262)
  Glucose, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Glucose, Day 14 | -0.033 (0.3197) | 0.057 (0.2787) | -0.109 (0.3220) | 0.046 (0.2481)
  Cholesterol, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Cholesterol, Day 8 | -0.148 (0.4156) | -0.116 (0.4323) | -0.054 (0.3518) | -0.201 (0.3767)
  Cholesterol, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Cholesterol, Day 9 | -0.036 (0.3198) | 0.005 (0.4131) | 0.081 (0.4041) | -0.186 (0.3427)
  Cholesterol, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Cholesterol, Day 14 | -0.102 (0.5090) | -0.181 (0.4539) | 0.032 (0.4605) | -0.273 (0.4303)
  Magnesium, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Magnesium, Day 8 | -0.017 (0.0443) | -0.018 (0.0379) | -0.011 (0.0364) | 0.005 (0.0394)
  Magnesium, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Magnesium, Day 9 | -0.020 (0.0389) | -0.001 (0.0370) | -0.013 (0.0200) | 0.009 (0.0328)
  Magnesium, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Magnesium, Day 14 | -0.013 (0.0431) | 0.002 (0.0334) | 0.008 (0.0379) | 0.003 (0.0353)
  Triglycerides, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Triglycerides, Day 8 | -0.019 (0.3330) | -0.111 (0.3637) | -0.002 (0.2699) | -0.100 (0.3027)
  Triglycerides, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Triglycerides, Day 9 | -0.050 (0.3006) | -0.097 (0.2744) | -0.153 (0.1572) | -0.151 (0.1979)
  Triglycerides, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Triglycerides, Day 14 | -0.052 (0.2523) | -0.127 (0.3297) | 0.031 (0.3383) | 0.035 (0.2705)
  Anion gap, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Anion gap, Day 8 | -0.2 (2.02) | 0.1 (1.35) | 0.0 (1.92) | -0.4 (2.10)
  Anion gap, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Anion gap, Day 9 | 0.8 (1.55) | 1.0 (1.10) | 1.2 (0.83) | 0.4 (1.65)
  Anion gap, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Anion gap, Day 14 | -0.4 (1.63) | -0.3 (1.51) | 0.1 (1.77) | -0.8 (1.75)
  Calcium, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Calcium, Day 8 | -0.059 (0.0737) | -0.037 (0.0795) | -0.034 (0.0744) | -0.063 (0.0617)
  Calcium, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Calcium, Day 9 | 0.001 (0.0798) | -0.025 (0.1053) | 0.050 (0.0825) | -0.032 (0.0780)
  Calcium, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Calcium, Day 14 | -0.010 (0.0754) | -0.003 (0.0555) | 0.042 (0.0671) | -0.020 (0.0584)
  Carbon dioxide, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Carbon dioxide, Day 8 | -1.0 (1.95) | -0.6 (1.62) | -1.2 (1.63) | -1.2 (2.12)
  Carbon dioxide, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Carbon dioxide, Day 9 | -0.5 (1.90) | -1.1 (1.45) | -0.8 (1.86) | -0.1 (1.10)
  Carbon dioxide, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Carbon dioxide, Day 14 | -0.2 (1.46) | 0.2 (1.92) | 0.1 (2.05) | 0.3 (1.79)
  Chloride, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Chloride, Day 8 | 0.7 (1.92) | -0.6 (1.62) | -0.2 (1.83) | -0.4 (2.03)
  Chloride, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Chloride, Day 9 | -0.6 (1.71) | -0.2 (1.40) | -1.0 (1.58) | -1.1 (2.28)
  Chloride, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Chloride, Day 14 | 1.0 (1.81) | 0.2 (1.85) | 0.5 (1.79) | 0.7 (2.22)
  Phosphate, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Phosphate, Day 8 | -0.009 (0.1060) | 0.031 (0.0971) | 0.018 (0.0966) | 0.004 (0.1388)
  Phosphate, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Phosphate, Day 9 | 0.016 (0.0819) | -0.001 (0.0641) | -0.016 (0.0985) | -0.005 (0.0593)
  Phosphate, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Phosphate, Day 14 | 0.027 (0.1225) | 0.000 (0.0961) | 0.054 (0.1156) | 0.047 (0.1375)
  Potassium, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Potassium, Day 8 | -0.02 (0.458) | -0.08 (0.302) | -0.12 (0.401) | -0.24 (0.455)
  Potassium, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Potassium, Day 9 | -0.05 (0.299) | -0.18 (0.343) | -0.03 (0.346) | -0.16 (0.295)
  Potassium, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Potassium, Day 14 | 0.07 (0.448) | 0.07 (0.373) | 0.12 (0.343) | 0.14 (0.393)
  Sodium, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Sodium, Day 8 | -0.4 (2.23) | -0.9 (1.96) | -0.9 (2.25) | -1.7 (1.68)
  Sodium, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Sodium, Day 9 | -0.4 (0.97) | -0.4 (1.12) | -0.4 (2.07) | -0.4 (2.01)
  Sodium, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Sodium, Day 14 | 0.5 (2.24) | -0.1 (1.87) | 0.8 (2.13) | 0.1 (2.12)
  Blood Urea Nitrogen, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Blood Urea Nitrogen, Day 8 | 0.751 (1.0248) | 0.890 (0.7840) | 0.385 (0.9919) | 0.225 (1.1465)
  Blood Urea Nitrogen, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Blood Urea Nitrogen, Day 9 | 0.557 (0.2739) | 0.631 (0.5449) | 0.154 (0.7635) | -0.060 (0.7601)
  Blood Urea Nitrogen, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Blood Urea Nitrogen, Day 14 | 0.098 (0.8195) | 0.173 (0.9149) | 0.008 (1.0030) | 0.010 (1.1314)

79. Secondary Outcome: Part 2: Change From Baseline in Chemistry Parameters: ALT, ALP, AST, GGT, Creatine Kinase, Lactate Dehydrogenase
Description: Blood samples were collected at indicated time points to analyze ALT, ALP, AST, GGT, creatine kinase, and lactate dehydrogenase. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visit. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
International units per liter
  ALT, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  ALT, Day 8 | -2.1 (4.76) | -0.9 (6.65) | -2.5 (4.90) | 2.0 (8.06)
  ALT, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  ALT, Day 9 | 0.7 (6.09) | -0.9 (2.34) | -0.6 (2.24) | 3.8 (9.87)
  ALT, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  ALT, Day 14 | -2.3 (5.67) | 0.6 (8.68) | -1.6 (6.24) | 1.7 (4.19)
  ALP, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  ALP, Day 8 | -2.2 (7.77) | -0.7 (4.55) | -1.2 (4.94) | -1.7 (4.71)
  ALP, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  ALP, Day 9 | -3.6 (7.29) | -0.1 (5.82) | 2.1 (5.84) | 1.1 (3.63)
  ALP, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  ALP, Day 14 | -1.8 (6.18) | -1.1 (7.33) | 0.5 (6.83) | -2.0 (6.55)
  AST, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  AST, Day 8 | -1.6 (3.66) | 0.0 (11.09) | -1.9 (2.49) | -0.2 (3.73)
  AST, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  AST, Day 9 | 0.9 (2.38) | -0.3 (1.62) | 0.7 (2.40) | 1.1 (3.98)
  AST, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  AST, Day 14 | -1.5 (3.42) | -0.7 (4.26) | -1.2 (3.36) | 0.0 (3.11)
  GGT, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  GGT, Day 8 | -0.5 (2.42) | -1.0 (2.44) | -0.7 (1.85) | -0.1 (3.51)
  GGT, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  GGT, Day 9 | -0.1 (1.97) | -0.4 (1.03) | 0.3 (1.22) | 0.3 (0.67)
  GGT, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  GGT, Day 14 | -1.0 (3.23) | -1.3 (2.74) | -0.8 (2.33) | -1.3 (4.28)
  Creatine kinase, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Creatine kinase, Day 8 | -18.9 (24.04) | 28.2 (446.48) | -31.7 (89.14) | -45.0 (97.35)
  Creatine kinase, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Creatine kinase, Day 9 | 39.7 (69.36) | -5.7 (18.29) | 63.9 (126.80) | 15.8 (29.26)
  Creatine kinase, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Creatine kinase, Day 14 | 8.8 (90.46) | -30.8 (80.07) | -22.5 (88.70) | -22.0 (100.57)
  Lactate dehydrogenase, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Lactate dehydrogenase, Day 8 | -11.2 (15.99) | -12.5 (20.51) | -11.9 (14.29) | -13.4 (17.89)
  Lactate dehydrogenase, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Lactate dehydrogenase, Day 9 | 1.9 (13.49) | -11.6 (12.66) | 0.0 (6.78) | 4.0 (9.72)
  Lactate dehydrogenase, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Lactate dehydrogenase, Day 14 | -5.4 (15.88) | -10.8 (20.17) | -3.3 (16.67) | -8.1 (15.00)

80. Secondary Outcome: Part 2: Change From Baseline in Chemistry Parameters: Creatinine, Urate, Total Bilirubin, Direct Bilirubin
Description: Blood samples were collected at indicated timepoints to analyze creatinine, urate, total bilirubin, and direct bilirubin. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visit. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Micromoles per liter
  Creatinine, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Creatinine, Day 8 | -0.03 (5.326) | 7.07 (7.515) | -1.15 (6.209) | 1.74 (5.394)
  Creatinine, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Creatinine, Day 9 | 1.59 (7.022) | 3.23 (4.312) | -0.48 (7.226) | 2.13 (6.927)
  Creatinine, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Creatinine, Day 14 | 0.67 (6.049) | 2.71 (5.478) | -0.37 (5.890) | 1.30 (4.255)
  Urate, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Urate, Day 8 | -6.0 (31.24) | 2.7 (23.18) | -8.1 (27.06) | -23.4 (26.58)
  Urate, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Urate, Day 9 | -4.7 (12.04) | 13.4 (24.46) | 17.7 (16.53) | -17.1 (24.15)
  Urate, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Urate, Day 14 | -4.1 (30.40) | -6.3 (28.01) | -4.6 (36.43) | -15.7 (26.94)
  Total Bilirubin, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Total Bilirubin, Day 8 | -2.15 (3.823) | -1.16 (2.946) | -0.17 (3.235) | -0.06 (3.984)
  Total Bilirubin, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Total Bilirubin, Day 9 | -0.52 (3.082) | 1.21 (2.806) | 1.10 (3.561) | -0.07 (2.873)
  Total Bilirubin, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Total Bilirubin, Day 14 | -0.65 (2.832) | 1.36 (3.546) | 1.54 (3.563) | 0.01 (3.193)
  Direct Bilirubin, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Direct Bilirubin, Day 8 | -0.33 (0.621) | -0.17 (0.581) | -0.06 (0.578) | 0.14 (0.821)
  Direct Bilirubin, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Direct Bilirubin, Day 9 | -0.12 (0.512) | 0.15 (0.589) | 0.19 (0.625) | 0.22 (0.503)
  Direct Bilirubin, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Direct Bilirubin, Day 14 | -0.12 (0.492) | 0.14 (0.582) | 0.19 (0.618) | 0.00 (0.582)

81. Secondary Outcome: Part 2: Change From Baseline in Chemistry Parameters: Albumin, Globulin, Total Protein
Description: Blood samples were collected at indicated timepoints to analyze albumin, globulin, and total protein. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visit. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Grams per liter
  Albumin, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Albumin, Day 8 | -2.5 (3.00) | -2.0 (2.58) | -1.6 (1.89) | -2.2 (2.05)
  Albumin, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Albumin, Day 9 | 0.4 (2.07) | -0.5 (3.14) | 1.1 (2.15) | 0.7 (2.45)
  Albumin, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Albumin, Day 14 | -0.9 (2.82) | -1.2 (2.32) | 0.1 (2.72) | -2.3 (2.21)
  Globulin, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Globulin, Day 8 | -0.6 (1.80) | -0.1 (1.96) | -0.2 (2.12) | -0.1 (1.96)
  Globulin, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Globulin, Day 9 | 0.0 (2.11) | -0.5 (2.38) | 0.4 (1.94) | 0.0 (1.63)
  Globulin, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Globulin, Day 14 | -0.4 (1.99) | 0.1 (1.88) | 0.6 (1.70) | -0.2 (1.46)
  Total protein, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Total protein, Day 8 | -3.1 (4.31) | -2.1 (3.86) | -1.8 (3.38) | -2.2 (3.45)
  Total protein, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Total protein, Day 9 | 0.4 (3.86) | -0.9 (5.19) | 1.6 (3.91) | 0.7 (3.95)
  Total protein, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Total protein, Day 14 | -1.3 (4.32) | -1.1 (3.41) | 0.7 (4.05) | -2.6 (2.98)

82. Secondary Outcome: Part 2: Change From Baseline in Chemistry Parameters: Amylase, Lipase
Description: Blood samples were collected at indicated timepoints to analyze amylase, lipase. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visit. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Units per liter
  Amylase, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Amylase, Day 8 | -0.8 (9.90) | -0.1 (11.55) | -3.6 (11.84) | -2.5 (10.69)
  Amylase, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Amylase, Day 9 | 3.1 (7.87) | 2.1 (7.61) | -1.0 (7.09) | 0.4 (2.84)
  Amylase, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Amylase, Day 14 | -2.3 (7.59) | -0.7 (9.91) | -4.1 (16.30) | -2.3 (11.00)
  Lipase, Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Lipase, Day 8 | 4.4 (27.20) | -0.7 (7.57) | -1.5 (9.36) | -3.0 (9.31)
  Lipase, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Lipase, Day 9 | 0.9 (3.63) | -0.9 (5.28) | 0.2 (5.52) | 1.7 (3.86)
  Lipase, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Lipase, Day 14 | -1.5 (5.66) | -0.5 (7.71) | -1.8 (8.08) | -2.6 (9.97)

83. Secondary Outcome: Part 2: Absolute Values for Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected at indicated time points to analyze the urine specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visit.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Ratio
  Baseline (Day -2) | 1.0152 (0.00779) | 1.0153 (0.00930) | 1.0167 (0.00894) | 1.0161 (0.00850)
  Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Day 8 | 1.0180 (0.00761) | 1.0164 (0.00846) | 1.0179 (0.00767) | 1.0188 (0.00590)
  Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Day 9 | 1.0189 (0.00973) | 1.0219 (0.00762) | 1.0179 (0.00595) | 1.0136 (0.00840)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Day 14 | 1.0165 (0.00779) | 1.0170 (0.00804) | 1.0165 (0.00782) | 1.0175 (0.00872)

84. Secondary Outcome: Part 2: Absolute Values for Urinalysis Parameter: pH
Description: Urine samples were collected at indicated time points to analyze the urine pH by dipstick test. The dipstick test gives results in a semi-quantitative manner indicating proportional concentrations in the urine sample. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0). Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visit.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
pH
  Baseline (Day -2) | 6.10 (0.386) | 6.19 (0.574) | 6.09 (0.479) | 6.13 (0.596)
  Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Day 8 | 5.90 (0.327) | 5.88 (0.415) | 5.98 (0.302) | 6.02 (0.278)
  Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Day 9 | 5.75 (0.264) | 5.91 (0.625) | 6.06 (0.527) | 6.20 (0.483)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Day 14 | 6.00 (0.491) | 6.00 (0.378) | 6.13 (0.447) | 6.12 (0.475)

85. Secondary Outcome: Part 2: Change From Baseline in Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected at indicated time points to analyze the urine specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visit. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Ratio
  Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Day 8 | 0.0034 (0.00849) | 0.0030 (0.00875) | 0.0019 (0.00727) | 0.0026 (0.01037)
  Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Day 9 | 0.0015 (0.00619) | 0.0015 (0.00708) | -0.0011 (0.01080) | -0.0020 (0.00850)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Day 14 | 0.0022 (0.00747) | 0.0037 (0.00838) | 0.0005 (0.00922) | 0.0016 (0.01055)

86. Secondary Outcome: Part 2: Change From Baseline in Urinalysis Parameter: pH
Description: Urine samples were collected at indicated time points to analyze the urine pH by dipstick test. The dipstick test gives results in a semi-quantitative manner indicating proportional concentrations in the urine sample. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0). Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visit. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -2), Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
pH
  Day 8: number analyzed (Participants) | 31 | 29 | 31 | 30
  Day 8 | -0.19 (0.441) | -0.33 (0.539) | -0.08 (0.389) | -0.18 (0.676)
  Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Day 9 | -0.35 (0.337) | -0.23 (0.344) | -0.11 (0.546) | 0.30 (0.350)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 29
  Day 14 | -0.13 (0.490) | -0.21 (0.590) | 0.06 (0.442) | -0.09 (0.708)

87. Secondary Outcome: Part 2: Number of Participants With Clinically Significant Abnormal 12-Lead ECG Findings
Description: as for outcome 35
Time Frame: Baseline(Day-2), Day1: 1 Hour, 2 Hours, 3 Hours, 4 Hours, 6 Hours; Day 2: 24 Hours, Day 4: 1 Hour, 2 Hours, 3 Hours, 4 Hours, 6 Hours, Day 5: 24 Hours; Day 7: 1 Hour, 2 Hours, 3 Hours, 4 Hours, 6 Hours; Day 8: 24 Hours; Day 9 and Day 14
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Participants
  Baseline (Day -2) | 0 | 0 | 0 | 0
  Day 1: 1 Hours | 0 | 0 | 0 | 0
  Day 1: 2 Hours | 0 | 0 | 0 | 0
  Day 1: 3 Hours | 0 | 0 | 0 | 0
  Day 1: 4 Hours | 0 | 0 | 0 | 0
  Day 1: 6 Hours | 0 | 0 | 0 | 0
  Day 2: 24 Hours | 0 | 0 | 0 | 0
  Day 4: 1 Hours | 0 | 0 | 0 | 0
  Day 4: 2 Hours | 0 | 0 | 0 | 0
  Day 4: 3 Hours | 0 | 0 | 0 | 0
  Day 4: 4 Hours | 0 | 0 | 0 | 0
  Day 4: 6 Hours | 0 | 0 | 0 | 0
  Day 5: 24 Hours | 0 | 0 | 0 | 0
  Day 7: 1 Hours | 0 | 0 | 0 | 0
  Day 7: 2 Hours | 0 | 0 | 0 | 0
  Day 7: 3 Hours | 0 | 0 | 0 | 0
  Day 7: 4 Hours | 0 | 0 | 0 | 0
  Day 7: 6 Hours | 0 | 0 | 0 | 0
  Day 8: 24 Hours | 0 | 0 | 0 | 0
  Day 9 | 0 | 0 | 0 | 0
  Day 14 | 0 | 0 | 0 | 0

88. Secondary Outcome: Part 2: Absolute Values for Vital Parameters: SBP and DBP
Description: SBP and DBP were measured in the semi-recumbent or supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Pre-dose, Day 1), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Millimeters of mercury
  SBP, Baseline (Pre-dose, Day 1) | 106.0 (9.39) | 106.7 (11.69) | 106.8 (9.03) | 105.4 (9.79)
  SBP, Day 2 | 103.9 (8.18) | 104.5 (9.05) | 105.6 (9.78) | 105.7 (10.10)
  SBP, Day 3 | 104.3 (9.82) | 103.8 (8.53) | 105.1 (9.41) | 105.3 (11.30)
  SBP, Day 4 | 103.1 (9.37) | 103.5 (11.25) | 105.3 (8.73) | 105.7 (10.05)
  SBP, Day 5 | 105.7 (9.50) | 103.3 (10.24) | 103.7 (8.65) | 106.8 (8.82)
  SBP, Day 6: number analyzed (Participants) | 41 | 40 | 40 | 40
  SBP, Day 6 | 105.2 (8.80) | 104.7 (8.60) | 105.7 (8.42) | 108.4 (9.44)
  SBP, Day 7: number analyzed (Participants) | 41 | 40 | 40 | 40
  SBP, Day 7 | 107.6 (10.34) | 106.7 (9.23) | 107.4 (8.68) | 107.4 (7.90)
  SBP, Day 8: number analyzed (Participants) | 41 | 40 | 40 | 40
  SBP, Day 8 | 109.9 (9.03) | 108.1 (9.40) | 109.4 (8.95) | 109.1 (9.24)
  ,SBP, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  ,SBP, Day 9 | 115.9 (9.72) | 104.2 (11.58) | 109.0 (7.48) | 105.8 (8.61)
  SBP, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 28
  SBP, Day 14 | 105.6 (9.51) | 108.0 (10.02) | 107.8 (9.38) | 106.3 (10.43)
  DBP, Baseline (Pre-dose, Day 1) | 61.1 (7.04) | 60.9 (6.61) | 62.1 (7.12) | 61.4 (6.18)
  DBP, Day 2 | 59.6 (6.27) | 59.3 (6.32) | 60.9 (6.65) | 60.9 (6.10)
  DBP, Day 3 | 60.9 (7.26) | 60.0 (7.46) | 61.0 (7.23) | 63.0 (7.80)
  DBP, Day 4 | 59.8 (7.61) | 60.0 (7.36) | 61.0 (5.40) | 62.8 (6.10)
  DBP, Day 5 | 60.3 (8.15) | 59.3 (6.23) | 59.1 (5.88) | 61.7 (5.44)
  DBP, Day 6: number analyzed (Participants) | 41 | 40 | 40 | 40
  DBP, Day 6 | 60.3 (5.69) | 60.1 (6.46) | 61.6 (6.99) | 62.4 (7.00)
  DBP, Day 7: number analyzed (Participants) | 41 | 40 | 40 | 40
  DBP, Day 7 | 61.0 (6.14) | 59.6 (6.89) | 61.1 (6.71) | 62.3 (6.28)
  DBP, Day 8: number analyzed (Participants) | 41 | 40 | 40 | 40
  DBP, Day 8 | 62.3 (6.72) | 62.6 (7.23) | 61.4 (7.18) | 62.7 (7.03)
  DBP, Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  DBP, Day 9 | 66.2 (5.67) | 56.6 (3.83) | 61.3 (5.41) | 65.8 (5.37)
  DBP, Day 14: number analyzed (Participants) | 30 | 29 | 31 | 28
  DBP, Day 14 | 61.6 (7.86) | 62.8 (6.65) | 61.8 (6.47) | 61.2 (6.91)

89. Secondary Outcome: Part 2: Absolute Values for Vital Parameter: Pulse Rate
Description: Pulse rate was measured in the semi-recumbent or supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Pre-dose, Day 1), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, and Day 14
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Beats per minute
  Baseline (Pre-dose, Day 1) | 62.5 (9.32) | 60.4 (7.68) | 61.8 (9.46) | 61.0 (6.85)
  Day 2 | 61.9 (8.37) | 62.4 (8.04) | 61.6 (7.22) | 63.2 (9.05)
  Day 3 | 63.4 (9.67) | 63.0 (6.76) | 62.2 (6.46) | 63.9 (7.81)
  Day 4 | 63.4 (8.59) | 63.0 (7.38) | 63.5 (7.88) | 64.5 (7.76)
  Day 5 | 64.4 (8.57) | 62.4 (7.52) | 63.3 (8.32) | 66.0 (7.08)
  Day 6: number analyzed (Participants) | 41 | 40 | 40 | 40
  Day 6 | 62.0 (6.87) | 63.0 (7.17) | 63.7 (8.89) | 66.5 (7.13)
  Day 7: number analyzed (Participants) | 41 | 40 | 40 | 40
  Day 7 | 63.4 (7.36) | 61.6 (6.77) | 62.7 (7.40) | 65.8 (7.40)
  Day 8: number analyzed (Participants) | 41 | 40 | 40 | 40
  Day 8 | 63.9 (8.98) | 63.9 (6.75) | 63.9 (7.21) | 65.7 (6.92)
  Day 9: number analyzed (Participants) | 10 | 11 | 9 | 10
  Day 9 | 69.2 (7.48) | 66.8 (8.89) | 70.3 (12.72) | 70.4 (10.19)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 28
  Day 14 | 63.6 (9.47) | 63.6 (8.18) | 63.6 (6.49) | 61.1 (7.33)

90. Secondary Outcome: Part 2: Absolute Values for Vital Parameter: Temperature
Description: Temperature was measured in the semi-recumbent or supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value for each period, including those from unscheduled visits.
Time Frame: Baseline (Pre-dose, Day 1), Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11, Day 12, Day 13, and Day 14
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
Number analyzed (Participants) | 42 | 40 | 40 | 40
Degrees Celsius
  Baseline (Pre-dose, Day 1) | 36.25 (0.304) | 36.28 (0.335) | 36.22 (0.379) | 36.32 (0.303)
  Day 1: number analyzed (Participants) | 30 | 29 | 31 | 30
  Day 1 | 36.14 (0.302) | 36.29 (0.313) | 36.25 (0.245) | 36.21 (0.378)
  Day 2 | 36.22 (0.333) | 36.17 (0.266) | 36.18 (0.309) | 36.18 (0.331)
  Day 3 | 36.20 (0.449) | 36.09 (0.283) | 36.14 (0.353) | 36.15 (0.344)
  Day 4 | 36.21 (0.378) | 36.13 (0.353) | 36.18 (0.288) | 36.23 (0.344)
  Day 5 | 36.26 (0.407) | 36.08 (0.326) | 36.16 (0.272) | 36.18 (0.289)
  Day 6: number analyzed (Participants) | 41 | 40 | 40 | 40
  Day 6 | 36.21 (0.364) | 36.21 (0.393) | 36.17 (0.320) | 36.16 (0.304)
  Day 7: number analyzed (Participants) | 41 | 40 | 40 | 40
  Day 7 | 36.20 (0.315) | 36.19 (0.303) | 36.22 (0.310) | 36.22 (0.305)
  Day 8: number analyzed (Participants) | 41 | 40 | 40 | 40
  Day 8 | 36.28 (0.368) | 36.25 (0.312) | 36.32 (0.344) | 36.34 (0.271)
  Day 9: number analyzed (Participants) | 38 | 38 | 38 | 38
  Day 9 | 36.16 (0.431) | 36.18 (0.363) | 36.23 (0.327) | 36.12 (0.349)
  Day 10: number analyzed (Participants) | 28 | 27 | 29 | 28
  Day 10 | 36.05 (0.353) | 36.10 (0.323) | 36.17 (0.296) | 36.13 (0.360)
  Day 11: number analyzed (Participants) | 28 | 27 | 29 | 28
  Day 11 | 36.05 (0.276) | 36.22 (0.333) | 36.28 (0.397) | 36.19 (0.327)
  Day 12: number analyzed (Participants) | 28 | 27 | 29 | 27
  Day 12 | 36.10 (0.350) | 36.14 (0.285) | 36.26 (0.333) | 36.07 (0.333)
  Day 13: number analyzed (Participants) | 27 | 27 | 29 | 28
  Day 13 | 36.12 (0.327) | 36.25 (0.314) | 36.20 (0.308) | 36.21 (0.397)
  Day 14: number analyzed (Participants) | 30 | 29 | 31 | 28
  Day 14 | 36.25 (0.261) | 36.31 (0.328) | 36.36 (0.224) | 36.31 (0.368)

91. Other Pre Specified Outcome: Part 2: Change From Baseline in QTcF - For Placebo and Moxifloxacin Arm
Description: as for outcome 42
Time Frame: Baseline (Pre-dose, Day 1), Day 7: Predose and 0.5, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 Hours post dose
Population: QT/QTc Population. Only those participants with data available at specified time points were analyzed.
Measure: Least Squares Mean (90% Confidence Interval); unit: Milliseconds
Arm/Group | Part 2: Placebo | Part 2: Moxifloxacin 400 mg
Number analyzed (Participants) | 40 | 40
Milliseconds
  Day 7, Predose: number analyzed (Participants) | 38 | 40
  Day 7, Predose | 2.7 [1.01 to 4.46] | 3.3 [1.61 to 5.01]
  Day7, 0.5 Hour Post-dose: number analyzed (Participants) | 40 | 39
  Day7, 0.5 Hour Post-dose | -1.9 [-3.75 to 0.02] | -2.1 [-3.98 to -0.19]
  Day 7, 1 Hour Post-dose: number analyzed (Participants) | 40 | 39
  Day 7, 1 Hour Post-dose | -0.3 [-2.22 to 1.68] | -1.1 [-3.04 to 0.88]
  Day 7, 2 Hour Post-dose: number analyzed (Participants) | 40 | 38
  Day 7, 2 Hour Post-dose | -3.9 [-6.09 to -1.76] | 1.7 [-0.53 to 3.85]
  Day 7, 3 Hour Post-dose: number analyzed (Participants) | 40 | 39
  Day 7, 3 Hour Post-dose | -4.3 [-6.48 to -2.18] | 3.6 [1.44 to 5.77]
  Day7, 3.5 Hour Post-dose: number analyzed (Participants) | 38 | 39
  Day7, 3.5 Hour Post-dose | -4.4 [-6.33 to -2.38] | 4.5 [2.55 to 6.50]
  Day7, 4 Hour Post-dose: number analyzed (Participants) | 39 | 39
  Day7, 4 Hour Post-dose | -3.0 [-4.88 to -1.14] | 5.6 [3.75 to 7.50]
  Day7, 4.5 Hour Post-dose: number analyzed (Participants) | 39 | 39
  Day7, 4.5 Hour Post-dose | -2.6 [-4.57 to -0.53] | 5.9 [3.83 to 7.87]
  Day7, 5 Hour Post-dose: number analyzed (Participants) | 38 | 38
  Day7, 5 Hour Post-dose | -1.3 [-3.19 to 0.64] | 6.9 [4.97 to 8.80]
  Day7, 6 Hour Post-dose: number analyzed (Participants) | 38 | 39
  Day7, 6 Hour Post-dose | -2.9 [-5.25 to -0.52] | 5.3 [2.98 to 7.69]
  Day7, 8 Hour Post-dose: number analyzed (Participants) | 37 | 39
  Day7, 8 Hour Post-dose | -7.7 [-9.67 to -5.70] | -0.8 [-2.72 to 1.21]
  Day7, 10 Hour Post-dose: number analyzed (Participants) | 38 | 39
  Day7, 10 Hour Post-dose | -4.2 [-6.05 to -2.40] | 2.6 [0.76 to 4.37]
  Day7, 12 Hour Post-dose: number analyzed (Participants) | 37 | 39
  Day7, 12 Hour Post-dose | -2.0 [-4.12 to 0.10] | 3.3 [1.19 to 5.33]
  Day7, 24 Hour Post-dose: number analyzed (Participants) | 38 | 39
  Day7, 24 Hour Post-dose | -0.6 [-2.57 to 1.39] | 6.2 [4.28 to 8.21]

ADVERSE EVENTS:
Time Frame: All-cause mortality, Serious adverse events (SAEs), and non-SAEs were collected up to Day 9 in Part 1 and up to Day 51 in Part 2 of the study
Description: All cause mortality, SAEs and non-SAEs were reported for the Safety Population which comprised of all randomized participants who received at least 1 dose of study intervention. AE data has been presented treatment-wise and part-wise.
Arm/Group | Part 1: Placebo | Part 1: GSK3640254 500 mg | Part 2: Placebo | Part 2: Moxifloxacin 400 mg | Part 2: GSK3640254 100 mg | Part 2: GSK3640254 500 mg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/6 | 0/42 | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/6 | 0/42 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 2/2 | 1/6 | 7/42 | 4/40 | 5/40 | 10/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=2) | Part 1: GSK3640254 500 mg (N=6) | Part 2: Placebo (N=42) | Part 2: Moxifloxacin 400 mg (N=40) | Part 2: GSK3640254 100 mg (N=40) | Part 2: GSK3640254 500 mg (N=40)
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 6
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Medical device site dermatitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Trichomoniasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT04563845/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT04563845/SAP_001.pdf